CLINICAL TRIAL: NCT00603525
Title: A Double-blind, Randomized, Placebo Controlled, Parallel Group, Multi-center, Phase III Trial of Ofatumumab Investigating Clinical Efficacy in Patients With Active Rheumatoid Arthritis Who Have Previously Had an Inadequate Response to One or More TNF Antagonist Therapies
Brief Title: Investigating Clinical Efficacy of Ofatumumab in Adult Rheumatoid Arthritis (RA) Patients Who Had an Inadequate Response to TNF-α Antagonist Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Ofatumumab IV trials in RA were prematurely terminated because GSK refocused clinical development of autoimmune indications on the subcutaneous delivery.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110634; GEN411 (Other: GENMAB)
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Results first posted 2011-11-28 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-04

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ofatumumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ofatumumab (Experimental): 1000 mL dilution of 35ml of ofatumumab in sterile, pyrogen free 0.9% NaCl. Each treatment cycle consisting of two IV infusion taken 14 days apart. A total of 8 infusion cycles given over a 144 week period
  Interventions: Drug: Ofatumumab
- 1000 ml Saline (Placebo Comparator): 1000 mL sterile, pyrogen free 0.9% NaCl. A treatment cycle consisting of two IV infusion taken 14 days apart. Only one placebo treatment cycle provided over a 24 week period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ofatumumab — 1000 mL dilution of 35ml of ofatumumab in sterile, pyrogen free 0.9% NaCl. Each treatment cycle consisting of two IV infusion taken 14 days apart. A total of 8 infusion cycles given over a 144 week period
  Arms: Ofatumumab
Drug: Placebo — 1000 mL sterile, pyrogen free 0.9% NaCl. A treatment cycle consisting of two IV infusion taken 14 days apart. Only one placebo treatment cycle provided over a 24 week period
  Arms: 1000 ml Saline

SUMMARY:
This is a phase III, double-blind, randomized, multicenter, and parallel group trial with a duration of 24 weeks, followed by a 120 week Open-label Period. The primary purpose of the study is to demonstrate the efficacy and safety of ofatumumab in reducing clinical signs and symptoms in adult RA patients who had an inadequate response to TNF-α antagonist therapy.

DETAILED DESCRIPTION:
This study consist of a double-blind, placebo controlled, and parallel group part with eligible patients enrolled into a 24 week Double-Blind Period, and randomized in a 1:1 ratio to receive either ofatumumab or placebo in addition to their background methotrexate treatment. Patients who complete the 24 week Double-blind Period without receiving rescue DMARD treatment will then be eligible to proceed into the 120 week Open-label Period to receive repeat treatment courses with ofatumumab. In the Open-label Period ofatumumab treatment courses will be given at individualized time intervals only if a clinical response has been achieved following the previous treatment course, and followed by a subsequent worsening in disease activity.

Patients who have completed the Open-label Period or have been withdrawn will then enter a maximum 2 year Follow-up Period, or until there B-cells return to normal or to baseline levels, whichever occurs earlier

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Active disease at the time of screening as defined by:

  ≥ 8 swollen joints (of 66 joints assessed) and ≥ 8 tender joints (of 68 joints assessed), C-Reactive Protein (CRP) ≥ 1.0 mg/dL or Erythrocyte Sedimentation Rate (ESR) ≥ 22 mm/hour, DAS28≥3.2 (based on ESR);
* Inadequate response to previous or current TNF-alpha antagonist treatment;
* Treatment with methotrexate (MTX), 7.5-25 mg/week, for at least 12 weeks and at a stable dose for at least 4 weeks.

Exclusion Criteria:

* Patients with a history of a rheumatic autoimmune disease other than RA or with significant systemic involvement secondary to RA;
* Previous exposure to biologic anti-rheumatic therapies, including investigational compounds;
* Exposure to TNF-alpha antagonist treatment < 12 weeks prior to visit 2;
* Chronic or ongoing active infectious disease requiring systemic treatment;
* Clinically significant cardiac disease; History of significant cerebrovascular disease;
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral psychiatric disease, or evidence of demyelinating disease;
* Known HIV positive; Serologic evidence of Hepatitis B infection; Positive test for Hepatitis C; Positive plasma / white cell JC Virus PCR;
* Serum IgG < lower limit of normal;
* Breast feeding women or women with a positive pregnancy test at screening;
* Current participation in any other interventional clinical study;
* Patients known or suspected of not being able to comply with a study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2008-01; Primary Completion 2011-03 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (52):
- Argentina (4):
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, San Miguel de Tucumán
- Denmark (2):
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Silkeborg
- France (6):
  - GSK Investigational Site, Amiens, Picardie
  - GSK Investigational Site, Cahors
  - GSK Investigational Site, Corbeil-Essonnes
  - GSK Investigational Site, Échirolles
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
- Germany (9):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin, State of Berlin
- Italy (8):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Telese Terme (BN), Campania
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Varese, Lombardy
  - GSK Investigational Site, Prato, Tuscany
  - GSK Investigational Site, Padua, Veneto
- Netherlands (3):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Zwolle
- Norway (4):
  - GSK Investigational Site, Haugesund
  - GSK Investigational Site, Levanger
  - GSK Investigational Site, Lillehammer
  - GSK Investigational Site, Trondheim
- GSK Investigational Site, Lima, Lima Province, Peru
- South Korea (2):
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Spain (6):
  - GSK Investigational Site, Getafe/Madrid
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Mérida (Badajoz)
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- Sweden (2):
  - GSK Investigational Site, Oskarström
  - GSK Investigational Site, Stockholm
- United Kingdom (5):
  - GSK Investigational Site, Wishaw, Lanarkshire
  - GSK Investigational Site, Newcastle, Northumberland
  - GSK Investigational Site, Cannock
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Leytonstone, London

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study OFA110634 is comprised of a 24-week Double-blind (DB) Period, followed by a 120-week Open-label (OL) Period. Participants who complete the OL Period, or who are withdrawn, enter a Follow-up (FU) period (anticipated to be approximately 2 years).
Groups:
- Placebo: Placebo was administered as two 1000 milliliter (ml) intravenous (IV) infusions, one at Day 0 and the other at Day 14, in addition to background methotrexate (MTX) treatment (7.5-25 milligrams [mg]/week [oral, intramuscular, or subcutaneous] for 24 weeks) in the DB Period.
- Ofatumumab: Ofatumumab 700 mg (35 ml) was administered as two 1000 ml IV infusions, one at Day 0 and the other at Day 14, in addition to background MTX treatment (7.5 to 25 mg/week [oral, intramuscular, or subcutaneous] for 24 weeks) in the DB Period. Participants completing the 24-week DB Period without receiving rescue disease-modifying anti-rheumatic drug treatment were eligible to proceed into the 120-week OL Period to receive repeat ofatumumab treatment courses (at individualized time intervals if a clinical response had been achieved after the previous treatment course).
- Placebo or OFA 700 mg: FU Period: Participants randomized to DB treatment who completed the OL Period, who did not enter the OL Period, who did not qualify for retreatment, or who were withdrawn were to be followed until the number of B-cells and circulating IgG had returned to normal (according to the central laboratory) or Baseline levels or for a maximum of 2 years from the last scheduled visit in the DB or OL Periods, whichever occurred earlier. No investigational product was administered in the Follow-up Period.
Period: DB Treatment Period (24 Weeks)
Arm/Group | Placebo | Ofatumumab | Placebo or OFA 700 mg: FU Period
Started | 84 | 85 | 0
Completed | 67 | 63 | 0
Not Completed | 17 | 22 | 0
Not completed — Adverse Event | 3 | 9 | 0
Not completed — Lack of Efficacy | 7 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Withdrawal by Subject | 5 | 6 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Participant Met Stopping Criteria | 0 | 1 | 0
Period: OL Treatment Period (120 Weeks)
Arm/Group | Placebo | Ofatumumab | Placebo or OFA 700 mg: FU Period
Started | 0 | 125 (61 participants received OFA during the DB Period; 64 received placebo during the DB Period.) | 0
Completed | 0 | 13 | 0
Not Completed | 0 | 112 | 0
Not completed — Adverse Event | 0 | 12 | 0
Not completed — Lack of Efficacy | 0 | 13 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Protocol-defined Stopping Criteria Met | 0 | 5 | 0
Not completed — Study Closed/Terminated | 0 | 71 | 0
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 8 | 0
Period: Follow-up Period (Approximately 2 Years)
Arm/Group | Placebo | Ofatumumab | Placebo or OFA 700 mg: FU Period
Started | 0 | 0 | 124 (124 participants (par) completing/withdrawing from the DB or OL Periods attended >=1 follow-up visit)
Unknown Reason for Withdrawal | 0 | 0 | 111 (As par. were not on active drug during the Follow-up Period, withdrawal reasons were not collected.)
Completed | 0 | 0 | 13
Not Completed | 0 | 0 | 111
Not completed — Unknown Reason for Withdrawal | 0 | 0 | 111

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo was administered as two 1000 milliliter (ml) intravenous (IV) infusions, one at Day 0 and the other at Day 14, in addition to background methotrexate (MTX) treatment (7.5 to 25 milligrams [mg]/week [oral, intramuscular, or subcutaneous] for 24 weeks).
- Ofatumumab 700 mg: Ofatumumab 700 mg (35 ml) was administered as two 1000 ml IV infusions, one at Day 0 and the other at Day 14, in addition to background MTX treatment (7.5 to 25 mg/week [oral, intramuscular, or subcutaneous] for 24 weeks).
- Total: Total of all reporting groups
Arm/Group | Placebo | Ofatumumab 700 mg | Total
Number analyzed (Participants) | 84 | 85 | 169
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.3 (11.69) | 53.7 (13.64) | 53.5 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 73 | 140
  Male | 17 | 12 | 29
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 35 | 35 | 70
  Not Hispanic/Latino | 49 | 50 | 99

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 20% Improvement From Baseline in Their American College of Rheumatology (ACR) Score (ACR20) at Week 24
Description: The ACR score was based on improvement from baseline in tender (TJC) and swollen joint counts (SJC). A participant had achieved ACR20 if he experienced >=20% improvement from baseline in TJC and SJC and a >=20% improvement from baseline in 3 out of 5 of the following assessments: participant pain assessment on a 100 millimeter (mm) visual analog scale (VAS), participant global assessment on a 100 mm VAS scale, physician global assessment on a 100 mm VAS scale, participant self-assessed disability, and C-reactive protein.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat (ITT) Population: all randomized participants who were exposed to investigational product irrespective of their compliance to the planned course of treatment. Participants were analyzed according to their randomized treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 84 | 85
participants | 16 | 36

2. Secondary Outcome: Number of Participants With a 20% Improvement From Baseline in Their American College of Rheumatology (ACR) Score (ACR20) at Weeks 4, 8, 12, 16, and 20
Description: as for outcome 1
Time Frame: Baseline and Weeks 4, 8, 12, 16, and 20
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 84 | 85
participants
  Week 4 | 22 | 25
  Week 8 | 23 | 29
  Week 12 | 30 | 36
  Week 16 | 23 | 36
  Week 20 | 21 | 40

3. Secondary Outcome: Number of Participants With a 50% Improvement From Baseline in Their ACR Score (ACR50) at Weeks 4, 8, 12, 16, 20, and 24
Description: The ACR score was based on improvement from baseline in tender (TJC) and swollen joint counts (SJC). A participant had achieved ACR50 if he experienced >=50% improvement from baseline in TJC and SJC and a >=50% improvement from baseline in 3 out of 5 of the following assessments: participant pain assessment on a 100 millimeter (mm) visual analog scale (VAS), participant global assessment on a 100 mm VAS scale, physician global assessment on a 100 mm VAS scale, participant self-assessed disability, and C-reactive protein.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 84 | 85
participants
  Week 4 | 9 | 4
  Week 8 | 8 | 9
  Week 12 | 11 | 17
  Week 16 | 10 | 17
  Week 20 | 8 | 18
  Week 24 | 5 | 19

4. Secondary Outcome: Number of Participants With a 70% Improvement From Baseline in Their ACR Score (ACR70) at Weeks 4, 8, 12, 16, 20, and 24
Description: The ACR score was based on improvement from baseline in tender (TJC) and swollen joint counts (SJC). A participant had achieved ACR70 if he experienced >=70% improvement from baseline in TJC and SJC and a >=70% improvement from baseline in 3 out of 5 of the following assessments: participant pain assessment on a 100 millimeter (mm) visual analog scale (VAS), participant global assessment on a 100 mm VAS scale, physician global assessment on a 100 mm VAS scale, participant self-assessed disability, and C-reactive protein.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 84 | 85
participants
  Week 4 | 3 | 0
  Week 8 | 2 | 3
  Week 12 | 3 | 5
  Week 16 | 3 | 5
  Week 20 | 3 | 5
  Week 24 | 3 | 6

5. Secondary Outcome: Mean Disease Activity Score Based on 28 Joints (DAS28) at Weeks 4, 8, 12, 16, 20, and 24 Using C-reactive Protein (CRP) as the Acute Phase Reactant (APR)
Description: The DAS28 is a clinical index of rheumatoid arthritis disease activity (DA) that combines information from swollen and tender joints (jts.), the APR, and general health (patient global assessment). The following jts. were assessed on both sides of the body: shoulder, elbow, wrist, metacarpophalangeal (5 per side), proximal interphalangeal (5 per side), and knee. The level of DA can be interpreted as low (DAS28<=3.2), moderate (3.2<DAS28<=5.1), or high (DAS28>5.1); total score, 0-9.4. A DAS28 <2.6 corresponds to remission. APRs are a class of proteins that are useful markers for inflammation.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population. Only those participants contributing values at the relevant visit were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 80 | 73
scores on a scale
  Week 4, n=80, 73 | 5.00 (1.492) | 5.02 (1.361)
  Week 8, n=74, 73 | 4.96 (1.352) | 4.60 (1.300)
  Week 12, n=73, 71 | 4.86 (1.537) | 4.16 (1.194)
  Week 16, n=69, 71 | 4.88 (1.526) | 4.17 (1.273)
  Week 20, n=67, 68 | 4.91 (1.505) | 4.04 (1.262)
  Week 24, n=68, 67 | 5.21 (1.324) | 4.22 (1.432)

6. Secondary Outcome: Change From Baseline in DAS28 at Weeks 4, 8, 12, 16, 20, and 24 Using CRP as the Acute Phase Reactant
Description: The DAS28 is a clinical index of rheumatoid arthritis disease activity (DA) that combines information from swollen and tender joints, the APR, and general health (patient global assessment). The level of DA can be interpreted as low (DAS28<=3.2), moderate (3.2<DAS28<=5.1), or high (DAS28>5.1); total score, 0-9.4. A DAS28 <2.6 corresponds to remission. APRs are a class of proteins that are useful markers for inflammation. Change from baseline in DAS28 is calculated as the Week 4, 8, 12, 16, 20, and 24 values minus the baseline value.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population. Only those participants contributing values at baseline and the relevant visit were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 80 | 73
scores on a scale
  Week 4, n=80, 73 | -0.83 (1.237) | -0.89 (1.094)
  Week 8, n=74, 73 | -0.81 (1.127) | -1.22 (1.142)
  Week 12, n=73, 71 | -0.92 (1.382) | -1.64 (1.242)
  Week 16, n=69, 71 | -0.86 (1.362) | -1.64 (1.318)
  Week 20, n=67, 68 | -0.79 (1.270) | -1.75 (1.311)
  Week 24, n=68, 67 | -0.51 (1.142) | -1.56 (1.370)

7. Secondary Outcome: Mean DAS28 at Weeks 4, 8, 12, 16, 20, and 24 Using Erythrocyte Sedimentation Rate (ESR) as the Acute Phase Reactant (ARP)
Description: as for outcome 5
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population. Only those participants contributing values at the relevant visit were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 80 | 74
scores on a scale
  Week 4, n=80, 74 | 5.84 (1.455) | 5.80 (1.390)
  Week 8, n=74, 72 | 5.76 (1.327) | 5.41 (1.335)
  Week 12, n=73, 71 | 5.60 (1.498) | 4.99 (1.269)
  Week 16, n=69, 71 | 5.66 (1.481) | 4.95 (1.356)
  Week 20, n=67, 68 | 5.74 (1.539) | 4.79 (1.312)
  Week 24, n=68, 67 | 5.96 (1.358) | 5.03 (1.537)

8. Secondary Outcome: Change From Baseline in DAS28 at Weeks 4, 8, 12, 16, 20, and 24 Using ESR as the Acute Phase Reactant
Description: as for outcome 6
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population. Only those participants contributing values at baseline and the relevant visit were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 80 | 74
scores on a scale
  Week 4, n=80, 74 | -0.85 (1.210) | -0.98 (1.105)
  Week 8, n=74, 72 | -0.88 (1.117) | -1.28 (1.165)
  Week 12, n=73, 71 | -1.05 (1.332) | -1.70 (1.304)
  Week 16, n=69, 71 | -0.95 (1.353) | -1.75 (1.350)
  Week 20, n=67, 68 | -0.85 (1.299) | -1.89 (1.299)
  Week 24, n=68, 67 | -0.63 (1.211) | -1.64 (1.473)

9. Secondary Outcome: Number of Participants With the Indicated European League Against Rheumatism (EULAR) Response at Weeks 4, 8, 12, 16, 20, and 24 Using CRP as the Acute Phase Reactant
Description: The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 <=3.2; moderate responders: change from baseline >1.2 with DAS28 <=3.2 to >5.1 or change from baseline >0.6 to <=1.2 with DAS28 <=3.2 to <=5.1); non-responders: change from baseline <=0.6 or change from baseline >0.6 and <=1.2 with DAS28 >5.1.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 84 | 85
participants
  Week 4, Good | 15 | 8
  Week 4, Moderate | 18 | 25
  Week 4, None | 47 | 40
  Week 8, Good | 11 | 11
  Week 8, Moderate | 23 | 31
  Week 8, None | 40 | 31
  Week 12, Good | 13 | 14
  Week 12, Moderate | 22 | 39
  Week 12, None | 38 | 18
  Week 16, Good | 9 | 17
  Week 16, Moderate | 23 | 33
  Week 16, None | 37 | 21
  Week 20, Good | 10 | 18
  Week 20, Moderate | 21 | 32
  Week 20, None | 36 | 18
  Week 24, Good | 6 | 15
  Week 24, Moderate | 19 | 29
  Week 24, None | 43 | 23

10. Secondary Outcome: Number of Participants With the Indicated European League Against Rheumatism (EULAR) Response at Weeks 4, 8, 12, 16, 20, and 24 Using ESR as the Acute Phase Reactant
Description: as for outcome 9
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 84 | 85
participants
  Week 4, Good | 3 | 4
  Week 4, Moderate | 29 | 21
  Week 4, None | 48 | 49
  Week 8, Good | 2 | 5
  Week 8, Moderate | 28 | 33
  Week 8, None | 44 | 34
  Week 12, Good | 2 | 7
  Week 12, Moderate | 36 | 41
  Week 12, None | 35 | 23
  Week 16, Good | 3 | 6
  Week 16, Moderate | 29 | 43
  Week 16, None | 37 | 22
  Week 20, Good | 1 | 5
  Week 20, Moderate | 27 | 46
  Week 20, None | 39 | 17
  Week 24, Good | 2 | 6
  Week 24, Moderate | 20 | 37
  Week 24, None | 46 | 24

11. Secondary Outcome: Median of the Largest Integer n, for Which a Participant Met the ACR Criteria Requiring an Improvement of n% (ACRn) at Weeks 4, 8, 12, 16, 20, and 24
Description: ACRn = the largest integer n for which a participant (par.) met the criteria requiring an improvement of n%. ACRn is a measure characterizing percentage (%) improvement from baseline (IFBL). A par. with an ACRn of X had an improvement of >=X% in tender/swollen joints (TJC/SJC), and an improvement of >=X% in 3 of the 5 parameters (patient [pt] pain assessment, pt global assessment [GA], physician GA, pt self-assessed disability, acute phase reactant). ACRn = min(TJC % IFBL, SJC % IFBL, composite measure % IFBL). Composite measure % IFBL is the 3rd highest value of % IFBL for the 5 parameters.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population. This trial was terminated prematurely due to the Sponsor's decision to not pursue clinical development of the IV formulation of ofatumumab in an autoimmune indication; thus, no participants were analyzed for this endpoint.
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Weeks 4, 8, 12, 16, 20, and 24
Description: The HAQ-DI is a 20-question instrument used to assess the degree of difficulty a participant had in accomplishing tasks in 8 functional areas (FAs): dressing, arising, eating, walking, hygiene, reaching, gripping, and errands/chores. Responses for each FA were scored from 0 (no difficulty) to 3 (inability to perform a task). The total score (range of 0-3) was calculated by adding the 8 individual FA scores, then dividing this sum by the total number of components answered. Responders were defined as participants achieving an improvement from baseline in the HAQ-DI score at Week 24 of >=0.22.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population. Only those participants contributing values at baseline and the relevant visit were analyzed.
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 75 | 72
scores on a scale
  Week 4, n=75, 72 | -0.13 [-1.9 to 0.8] | -0.13 [-1.9 to 1.4]
  Week 8, n=69, 68 | -0.25 [-2.1 to 1.1] | -0.38 [-1.6 to 0.9]
  Week 12, n=68, 65 | -0.13 [-2.3 to 1.0] | -0.38 [-1.9 to 1.0]
  Week 16, n=65, 64 | -0.13 [-2.1 to 1.0] | -0.38 [-2.0 to 0.5]
  Week 20, n=64, 64 | -0.13 [-2.3 to 1.1] | -0.38 [-2.1 to 1.3]
  Week 24, n=63, 61 | 0.00 [-2.3 to 1.0] | -0.38 [-2.1 to 1.5]

13. Secondary Outcome: Change From Baseline in Tender Joint Count at Week 24
Description: Change from baseline in tender joint count was calculated as the Week 24 count minus the baseline count. A total of 68 joints were assessed. Joints were classified as either tender or not tender by an independent assessor, who had documented experience in performing joint assessments.
Time Frame: Baseline and Week 24
Population: ITT Population. Only those participants contributing values at baseline and the relevant visit were analyzed.
Measure: Median (Full Range); unit: tender joints
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 68 | 66
tender joints | -5 [-46 to 23] | -11 [-56 to 14]

14. Secondary Outcome: Change From Baseline in Swollen Joint Count at Week 24
Description: Change from baseline in swollen joint count was calculated as the Week 24 count minus the baseline count. A total of 66 joints were assessed. Joints were classified as either swollen or not swollen by an independent assessor, who had documented experience in performing joint assessments.
Time Frame: Baseline and Week 24
Population: ITT Population. Only those participants contributing values at baseline and the relevant visit were analyzed.
Measure: Median (Full Range); unit: swollen joints
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 68 | 66
swollen joints | -3.50 [-27 to 37] | -7.50 [-27 to 33]

15. Secondary Outcome: Change From Baseline in CRP at Week 24
Description: Blood samples for the determination of CRP were taken at pre-specified visits and were sent to the central laboratory for analysis. Change from baseline in CRP was calculated as the Week 24 value minus the baseline value. CRP is an acute-phase protein whose plasma concentration increases in response to inflammation. CRP is a useful marker of inflammation.
Time Frame: Baseline and Week 24
Population: ITT Population. Only those participants contributing values at baseline and the relevant visit were analyzed.
Measure: Median (Full Range); unit: milligrams per liter (mg/L)
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 66 | 66
milligrams per liter (mg/L) | 1.05 [-51.5 to 94.0] | -2.85 [-150.6 to 41.4]

16. Secondary Outcome: Change From Baseline in ESR at Week 24
Description: ESR is measured by a blood test that shows the rate at which red blood cells sediment in a period of 1 hour. Blood samples for the determination of ESR were taken at pre-specified visits and were measured immediately at the trial site. Change from baseline in ESR was calculated as the Week 24 value minus the baseline value.
Time Frame: Baseline and Week 24
Population: ITT Population. Only those participants contributing values at baseline and the relevant visit were analyzed.
Measure: Median (Full Range); unit: millimeters per hour (mm/hr)
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 67 | 67
millimeters per hour (mm/hr) | 0.00 [-73 to 52] | -12.00 [-100 to 45]

17. Secondary Outcome: Change From Baseline in the Participant-assessed Pain Score Using Visual Analogue Scale (VAS) at Week 24
Description: A horizontal VAS of 100 mm was used to report the participant's level of joint pain. The scale ranged from 0 (no pain) to 100 (unbearable pain). Participants were instructed to draw a vertical line through the horizontal line to indicate how much joint pain they had. The distance from the "no pain" end to the vertical line drawn by the participant was the joint pain score. Change from baseline was calculated as the Week 24 value minus the baseline value.
Time Frame: Baseline and Week 24
Population: as for outcome 11
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Change From Baseline in Participant-assessed Global Disease Score Using VAS at Week 24
Description: The participant used a horizontal VAS of 100 mm for overall assessment of disease. The scale ranged from 0 (very well) to 100 (very poor). Participants were instructed to draw a vertical line through the horizontal line to indicate the state of the arthritis. The distance from the "very well" end to the vertical line drawn by the participant was the global disease assessment score. Change from baseline in participant-assessed global disease was calculated as the Week 24 value minus the baseline value.
Time Frame: Baseline and Week 24
Population: as for outcome 11
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Change From Baseline in the Physician-assessed Global Disease Score Using VAS at Week 24
Description: The physician used a horizontal VAS of 100 mm for overall assessment of disease. The scale ranged from 0 (very well) to 100 (very poor). Physicians were instructed to draw a vertical line through the horizontal line to indicate the state of the arthritis. The distance from the "very well" end to the vertical line drawn by the participant was the global disease assessment score. Change from baseline in the physician-assessed global disease was calculated as the Week 24 value minus the baseline value.
Time Frame: Baseline and Week 24
Population: as for outcome 11
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy (FACIT) Questionnaire Score at Week 24
Description: The FACIT-F score has a valid range of values from 0 to 52, with a higher score indicating a lower burden of fatigue. The subset determining fatigue contains 13 questions. Responses to each question were scored from 0, indicating "Not at all fatigued," to 4, indicating "Very much fatigued."
Time Frame: Baseline and Week 24
Population: as for outcome 11
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Change From Baseline in the Short-Form 36 (SF-36v2) Norm-based Scores for Physical Component Summary and Physical Items at Week 24
Description: The SF-36v2 is a standardized questionnaire used to measure overall subjective health status by measuring 8 health-related parameters (each scored from 0 [poorer health] to 100 [better health]): body pain, general mental health (MH), perception of general health, physical functioning, role limitations (RL) caused by mental condition, RL caused by a physical condition, social functioning, and vitality. It yields an 8-scale profile of functional health and well-being scores, as well as psychometrically based physical and MH summary measures and a preference-based health utility index.
Time Frame: Baseline and Week 24
Population: as for outcome 11
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Change From Baseline in the SF-36v2 Norm-based Scores for Mental Component Summary and Mental Items at Week 24
Description: The SF-36v2 is a standardized questionnaire used to measure overall subjective health status by measuring 8 health-related parameters (each scored from 0 [poorer health] to 100 [better health]): body pain, general mental health (MH), perception of general health, physical functioning, role limitations (RL) caused by mental condition, RL caused by a physical condition, social functioning, and vitality. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and MH summary measures and a preference-based health utility index.
Time Frame: Baseline and Week 24
Population: as for outcome 11
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Biomarker Levels for Anti-CCP, RF-IgA, RF-IgG, and RF-IgM at Baseline and Week 4
Description: The following biomarkers were assessed: Anti-Cyclic Citrullinated Peptide 3 antibody (Anti-CCP), Rheumatoid factor IgA (RF-IgA), RF IgG (RF-IgG), and RF IgM (RF-IgM). Measurements of RF were used to characterize participants' disease activity and immune status. Anti-CCP was used to characterize the disease type and the immune status of the participants. Assessments for which results were below the lower limit of quantification (LLQ) were reported using a value of LLQ/2. Assessments for which results were above the upper limit of quantification (ULQ) were reported using a value of ULQ.
Time Frame: Baseline and Week 4
Population: ITT Population. Only those participants contributing values at the relevant visit were analyzed.
Measure: Median (Full Range); unit: Units/Liter
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 81 | 82
Units/Liter
  Anti-CCP, Baseline, n=81, 82 | 466 [8 to 10828] | 449.5 [8 to 8261]
  RF-IgA, Baseline, n=81, 81 | 9 [2.5 to 100] | 11 [2.5 to 100]
  RF-IgA, Week 4, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | 100 [100 to 100]
  IgG, Baseline, n=81, 81 | 5 [2.5 to 100] | 2.5 [2.5 to 100]
  IgG, Week4, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | 5 [5 to 5]
  RF-IgM, Baseline, n=81, 81 | 92 [2.5 to 100] | 68 [2.5 to 100]
  RF-IgM, Week 4, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | 43 [43 to 43]

24. Secondary Outcome: Number of Participants With Positive Human Anti-human Antibodies (HAHA) at Week 24
Description: Detection of human anti-human antibodies (HAHAs) against ofatumumab was to be performed by Electrochemiluminescent (ECL) Meso-Scale Discovery (MSD) immunoassay. Positive samples from the binding antibody test were also tested in a neutralizing antibody assay.
Time Frame: Baseline and Week 24
Population: as for outcome 11
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Change From Baseline in Levels of IgA, IgG and IgM at Week 12 and Week 24
Description: The following immunoglobulins were assessed: IgA, IgG and IgM. Immunoglobulins, or antibodies, are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Low levels indicate immuno-suppression.
Time Frame: Baseline, Week 12, and Week 24
Population: Safety Population: identical to the ITT population except that participants were analyzed according to their actual treatment when this differed from their randomized treatment. Only those participants contributing values at baseline and the relevant visit were analzyed.
Measure: Median (Full Range); unit: grams per Liter (g/L)
Groups:
- Placebo: Placebo was administered as two 1000 ml IV infusions, one at Day 0 and the other at Day 14, in addition to background MTX treatment (7.5 to 25 mg/week [oral, intramuscular, or subcutaneous] for 24 weeks).
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 79 | 75
grams per Liter (g/L)
  IgA, Week 12; n=79, 75 | -0.020 [-1.72 to 1.47] | -0.250 [-2.32 to 0.65]
  IgA, Week 24; n=69, 68 | 0.050 [-1.51 to 1.47] | -0.350 [-2.58 to 0.81]
  IgG, Week 12; n=79, 75 | -0.400 [-7.30 to 7.20] | -1.300 [-7.60 to 2.10]
  IgG, Week 24; n=69, 68 | -0.700 [-8.30 to 8.30] | -1.615 [-9.70 to 4.80]
  IgM, Week 12; n=79, 75 | -0.040 [-1.58 to 0.75] | -0.260 [-2.92 to 0.17]
  IgM, Week 24; n=69, 68 | -0.050 [-1.30 to 1.47] | -0.355 [-4.12 to 0.40]

26. Secondary Outcome: Minimum DAS28-ESR Score During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The DAS28 is a clinical index of rheumatoid arthritis disease activity that combines information from swollen and tender joints (jts.), the APR, and general health (patient global assessment). The following jts. were assessed on both sides of the body: shoulder, elbow, wrist, metacarpophalangeal (5 per side), proximal interphalangeal (5 per side), and knee. The level of disease activity can be interpreted as low (DAS28<=3.2), moderate (3.2<DAS28<=5.1), or high (DAS28>5.1); total score, 0-9.4. A DAS28 <2.6 corresponds to remission. The values summarized are the minimum DAS28 score (i.e. lowest level of disease activity) achieved by each participant within the first 24 weeks of each treatment course (TC), assessed using erythrocyte sedimentation rate (ESR; rate at which red blood cells sediment in 1 hour).
Time Frame: First 24 weeks of each treatment course (assessed up to Week 144)
Population: As Treated (AT) Population: all participants who received at least one infusion of ofatumumab in the DB and/or OL Period
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 148 | 0
Scores on a scale
  TC 1, n=0, 148, 0 |  | 4.64 (1.511) |
  TC 2, n=0, 92, 0 |  | 4.08 (1.129) |
  TC 3, n=0, 62, 0 |  | 4.09 (1.346) |
  TC 4, n=0, 29, 0 |  | 3.84 (1.437) |
  TC 5, n=0, 13, 0 |  | 3.95 (1.327) |
  TC 6, n=0, 6, 0 |  | 3.33 (1.245) |

27. Secondary Outcome: Minimum DAS28-CRP Score During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The DAS28 is a clinical index of rheumatoid arthritis disease activity that combines information from swollen and tender joints (jts.), the APR, and general health (patient global assessment). The following jts. were assessed on both sides of the body: shoulder, elbow, wrist, metacarpophalangeal (5 per side), proximal interphalangeal (5 per side), and knee. The level of disease activity can be interpreted as low (DAS28<=3.2), moderate (3.2<DAS28<=5.1), or high (DAS28>5.1); total score, 0-9.4. A DAS28 <2.6 corresponds to remission. The values summarized are the minimum DAS28 score (i.e. lowest level of disease activity) achieved by each participant within the first 24 weeks of each treatment course, assessed using C-reactive Protein (CRP: used to monitor acute inflammatory phases of rheumatoid arthritis).
Time Frame: First 24 weeks of each treatment course (assessed up to Week 144)
Population: AT Population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 147 | 0
scores on a scale
  TC 1, n=0, 147, 0 |  | 3.86 (1.443) |
  TC 2, n=0, 92, 0 |  | 3.37 (1.120) |
  TC 3, n=0, 62, 0 |  | 3.35 (1.181) |
  TC 4, n=0, 29, 0 |  | 3.15 (1.214) |
  TC 5, n=0, 13, 0 |  | 3.23 (1.129) |
  TC 6, n=0, 6, 0 |  | 2.84 (1.193) |

28. Secondary Outcome: Minimum Change From Baseline DAS28-ESR Score, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The level of rheumatoid arthritis disease activity based on the DAS28 score is defined as low if DAS28 <=3.2, moderate if 3.2< DAS28 <=5.1, or high if DAS28 > 5.1. A DAS28 <2.6 corresponds to clinical remission. The values summarized are the minimum change from baseline DAS28 score (i.e. greatest change in disease activity during the treatment course) achieved by each participant within the first 24 weeks of each treatment course, assessed by using ESR. Baseline score was determined at the start of each treatment course. For change from baseline, participants had to have both a baseline DAS28 value for the treatment course (i.e., the latest value on or before the date of infusion A of the treatment course, providing it was done within a 14 day window prior to the date of infusion A) and a DAS28 value during the treatment course (i.e., during first 24 weeks of each treatment course). Change from baseline was calculated as the value during the treatment course minus the baseline value.
Time Frame: First 24 weeks of each treatment course (assessed up to Week 144)
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 134 | 0
scores on a scale
  TC 1, n=0, 134, 0 |  | -2.04 (1.348) |
  TC 2, n=0, 90, 0 |  | -1.70 (1.090) |
  TC 3, n=0, 59, 0 |  | -1.52 (1.052) |
  TC 4, n=0, 28, 0 |  | -1.76 (1.499) |
  TC 5, n=0, 12, 0 |  | -1.50 (1.052) |
  TC 6, n=0, 6, 0 |  | -2.39 (0.581) |

29. Secondary Outcome: Minimum Change From Baseline DAS28-CRP Score, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The level of rheumatoid arthritis disease activity based on the DAS28 score is defined as low if DAS28 <=3.2, moderate if 3.2< DAS28 <=5.1, or high if DAS28 > 5.1. A DAS28 <2.6 corresponds to clinical remission. The values summarized are the minimum change from baseline DAS28 score (i.e. greatest change in disease activity during the treatment course) achieved by each participant within the first 24 weeks of each treatment course, assessed by using CRP. Baseline score was determined at the start of each treatment course. For change from baseline, participants had to have both a baseline DAS28 value for the treatment course (i.e., the latest value on or before the date of infusion A of the treatment course, providing it was done within a 14 day window prior to the date of infusion A) and a DAS28 value during the treatment course (i.e., during first 24 weeks of each treatment course). Change from baseline was calculated as the value during the treatment course minus the baseline value.
Time Frame: First 24 weeks of each treatment course (assessed up to Week 144)
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 134 | 0
scores on a scale
  TC 1, n=0, 134, 0 |  | -1.93 (1.297) |
  TC 2, n=0, 92, 0 |  | -1.65 (1.086) |
  TC 3, n=0, 61, 0 |  | -1.44 (1.006) |
  TC 4, n=0, 28, 0 |  | -1.65 (1.378) |
  TC 5, n=0, 12, 0 |  | -1.46 (1.006) |
  TC 6, n=0, 6, 0 |  | -2.20 (0.610) |

30. Secondary Outcome: Time to Retreatment, by Ofatumumab Treatment Course
Description: Time to retreatment is defined as the time in days between infusion A of each treatment course and infusion A of the following treatment course. For participants randomized to ofatumumab in the Double-blind Period, Treatment Course 1 refers to the course of ofatumumab received in the Double-blind Period. The minimum period allowed per protocol before retreatment was 24 weeks (end of Double-blind Period). For participants randomized to placebo in the Double-blind Period, Treatment Course 1 refers to the first course of ofatumumab received in the Open-label Period. The minimum period allowed per protocol before retreatment during the Open-label Period was 16 weeks.
Time Frame: From Baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 93 | 0
Days
  TC 1, n=0, 93, 0 |  | 32.79 (12.031) |
  TC 2, n=0, 63, 0 |  | 28.62 (11.108) |
  TC 3, n=0, 30, 0 |  | 24.56 (8.127) |
  TC 4, n=0, 13, 0 |  | 23.93 (6.143) |
  TC 5, n=0, 6, 0 |  | 19.07 (2.795) |
  TC 6, n=0, 0, 0 |  | NA (NA) — No participants were analyzed in this treatment group for Treatment Course 6. |

31. Secondary Outcome: Number of Participants Who Achieved Remission or Low Disease Activity Based on DAS28 (Using ESR), During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The DAS28 is a clinical index of rheumatoid arthritis disease activity that combines information from swollen and tender joints (jts.), the APR, and general health (patient global assessment). The following jts. were assessed on both sides of the body: shoulder, elbow, wrist, metacarpophalangeal (5 per side), proximal interphalangeal (5 per side), and knee. The level of disease activity can be interpreted as low (DAS28<=3.2), moderate (3.2<DAS28<=5.1), or high (DAS28>5.1); total score, 0-9.4. A DAS28 <2.6 corresponds to remission. Remission is defined as a DAS28 score <2.6 at any time during the first 24 weeks of each treatment course. Low disease activity is defined as a DAS28 score >=2.6 and <3.2 at any time during the first 24 weeks of each treatment course.
Time Frame: First 24 weeks of each treatment course (assessed up to Week 144)
Population: AT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 148 | 0
participants
  TC 1, Remission, n=0, 148, 0 |  | 15 |
  TC 1, Low Disease Activity, n=0, 148 |  | 7 |
  TC 2, Remission, n=0, 93, 0 |  | 5 |
  TC 2, Low Disease Activity, n=0, 93, 0 |  | 20 |
  TC 3, Remission, n=0, 63, 0 |  | 8 |
  TC 3, Low Disease Activity, n=0, 63, 0 |  | 8 |
  TC 4, Remission, n=0, 30, 0 |  | 6 |
  TC 4, Low Disease Activity, n=0, 30, 0 |  | 5 |
  TC 5, Remission, n=0, 13, 0 |  | 2 |
  TC 5, Low Disease Activity, n=0, 13, 0 |  | 2 |
  TC 6, Remission, n=0, 6, 0 |  | 2 |
  TC 6, Low Disease Activity, n=0, 6, 0 |  | 2 |

32. Secondary Outcome: Number of Participants Who Achieved Remission or Low Disease Activity Based on DAS28 (Using CRP), During the DB and OL Periods, by Ofatumumab Treatment Course
Description: as for outcome 31
Time Frame: First 24 weeks of each treatment course (assessed up to Week 144)
Population: AT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 148 | 0
participants
  TC 1, Remission, n=0, 148, 0 |  | 27 |
  TC 1, Low Disease Activity, n=0, 148, 0 |  | 26 |
  TC 2, Remission, n=0, 93, 0 |  | 24 |
  TC 2, Low Disease Activity, n=0, 93, 0 |  | 17 |
  TC 3, Remission, n=0, 63, 0 |  | 19 |
  TC 3, Low Disease Activity, n=0, 63, 0 |  | 10 |
  TC 4, Remission, n=0, 30, 0 |  | 10 |
  TC 4, Low Disease Activity, n=0, 30, 0 |  | 5 |
  TC 5, Remission,n=0, 13, 0 |  | 5 |
  TC 5, Low Disease Activity,n=0, 13, 0 |  | 1 |
  TC 6, Remission,n=0, 6, 0 |  | 3 |
  TC 6, Low Disease Activity,n=0, 6, 0 |  | 2 |

33. Secondary Outcome: Number of Participants With Any On-treatment Adverse Event or Serious Adverse Event, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; or is a congenital anomaly/birth defect. Medical or scientific judgment should have been exercised in other situations. Refer to the general AE/SAE module for a list of AEs (occurring at a frequency threshold >=2%) and SAEs.
Time Frame: First treatment (Day 0) until the participant terminated the trial, assessed up to Week 144
Population: AT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 148 | 0
Participants
  Any AE, TC 1, n=0, 148, 0 |  | 126 |
  Any AE, TC 2, n=0, 93, 0 |  | 60 |
  Any AE, TC 3, n=0, 63, 0 |  | 36 |
  Any AE, TC 4, n=0, 30, 0 |  | 17 |
  Any AE, TC 5, n=0, 13, 0 |  | 8 |
  Any AE, TC 6, n=0, 6, 0 |  | 5 |
  Any SAE, TC 1, n=0, 148, 0 |  | 20 |
  Any SAE, TC 2, n=0, 93, 0 |  | 10 |
  Any SAE, TC 3, n=0, 63, 0 |  | 2 |
  Any SAE, TC 4, n=0, 30, 0 |  | 0 |
  Any SAE, TC 5, n=0, 13, 0 |  | 0 |
  Any SAE, TC 6, n=0, 6, 0 |  | 0 |

34. Secondary Outcome: Number of Participants With the Indicated Electrocardiogram (ECG) Findings, During the OL Period
Description: The number of participants with normal, abnormal clinically significant (CS), and abnormal not clinically significant (NCS) ECG findings, as well as the number of participants with no results (NR), during the OL Period are presented. An overall interpretation of the ECG was made by the investigator, or the investigator could delegate this task to a cardiologist, if applicable.
Time Frame: From DB Period completion (Week 24) until the completion of the OL Period, assessed up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 117 | 0
Participants
  Week 48, normal, n=0, 117, 0 |  | 81 |
  Week 48, abnormal CS, n=0, 117, 0 |  | 0 |
  Week 48, abnormal NCS, n=0, 117, 0 |  | 34 |
  Week 48, NR, n=0, 117, 0 |  | 2 |
  Week 72, normal, n=0, 87, 0 |  | 59 |
  Week 72, abnormal CS, n=0, 87, 0 |  | 0 |
  Week 72, abnormal NCS, n=0, 87, 0 |  | 25 |
  Week 72, NR, n=0, 87, 0 |  | 3 |
  Week 96, normal, n=0, 57, 0 |  | 40 |
  Week 96, abnormal CS, n=0, 57, 0 |  | 0 |
  Week 96, abnormal NCS, n=0, 57, 0 |  | 16 |
  Week 96, NR, n=0, 57, 0 |  | 1 |
  Week 120, normal, n=0, 33, 0 |  | 16 |
  Week 120, abnormal CS, n=0, 33, 0 |  | 0 |
  Week 120, abnormal NCS, n=0, 33, 0 |  | 17 |
  Week 120, NR, n=0, 33, 0 |  | 0 |
  Week 144, normal, n=0, 17, 0 |  | 10 |
  Week 144, abnormal CS, n=0, 17, 0 |  | 0 |
  Week 144, abnormal NCS, n=0, 17, 0 |  | 7 |
  Week 144, NR, n=0, 17, 0 |  | 0 |

35. Secondary Outcome: Number of Participants With a CD19+ Cell Count Greater Than or Equal to the Lower Limit of Normal or the Baseline Value at Indicated the Time Point, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The number of participants with a CD19+ cell count greater than or equal to the lower limit of normal (LLN; reference range 0.11 to 0.66 giga [10^9] per liter) or the baseline value (whichever was lower) is presented. The baseline assessment is defined as the start of the Double-blind Period.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 136 | 0
Participants
  TC 1, Week 8, n=0, 136, 0 |  | 0 |
  TC 1, Week 16, n=0, 100, 0 |  | 0 |
  TC 1, Week 24, n=0, 99, 0 |  | 2 |
  TC 1, Week 32, n=0, 50, 0 |  | 1 |
  TC 1, Week 40, n=0, 30, 0 |  | 3 |
  TC 1, Week 48, n=0, 23, 0 |  | 1 |
  TC 1, Week 56, n=0, 14, 0 |  | 3 |
  TC 1, Week 64, n=0, 7, 0 |  | 1 |
  TC 1, Week 72, n=0, 4, 0 |  | 0 |
  TC 1, Week 80, n=0, 1, 0 |  | 0 |
  TC 1, Week 88, n=0, 1, 0 |  | 0 |
  TC 1, Week 96, n=0, 1, 0 |  | 0 |
  TC 1, Week 104, n=0, 2, 0 |  | 1 |
  TC 1, Week 112, n=0, 1, 0 |  | 0 |
  TC 1, Week 120, n=0, 1, 0 |  | 0 |
  TC 1, Week 128, n=0, 1, 0 |  | 0 |
  TC 1, Week 144, n=0, 1, 0 |  | 0 |
  TC 2, Week 8, n=0, 93, 0 |  | 0 |
  TC 2, Week 16, n=0, 80, 0 |  | 1 |
  TC 2, Week 24, n=0, 70, 0 |  | 0 |
  TC 2, Week 32, n=0, 31, 0 |  | 2 |
  TC 2, Week 40, n=0, 20, 0 |  | 2 |
  TC 2, Week 48, n=0, 11, 0 |  | 1 |
  TC 2, Week 56, n=0, 8, 0 |  | 0 |
  TC 2, Week 64, n=0, 6, 0 |  | 1 |
  TC 2, Week 72, n=0, 2, 0 |  | 0 |
  TC 2, Week 80, n=0, 2, 0 |  | 0 |
  TC 2, Week 96, n=0, 1, 0 |  | 0 |
  TC 3, Week 8, n=0, 60, 0 |  | 0 |
  TC 3, Week 16, n=0, 45, 0 |  | 0 |
  TC 3, Week 24, n=0, 29, 0 |  | 0 |
  TC 3, Week 32, n=0, 12, 0 |  | 1 |
  TC 3, Week 40, n=0, 4, 0 |  | 0 |
  TC 3, Week 48, n=0, 2, 0 |  | 1 |
  TC 3, Week 56, n=0, 1, 0 |  | 1 |
  TC 4, Week 8, n=0, 29, 0 |  | 0 |
  TC 4, Week 16, n=0, 24, 0 |  | 0 |
  TC 4, Week 24, n=0, 13, 0 |  | 0 |
  TC 4, Week 32, n=0, 4, 0 |  | 0 |
  TC 4, Week 40, n=0, 1, 0 |  | 0 |
  TC 4, Week 48, n=0, 1, 0 |  | 0 |
  TC 5, Week 8, n=0, 13, 0 |  | 0 |
  TC 5, Week 16, n=0, 8, 0 |  | 0 |
  TC 5, Week 24, n=0, 5, 0 |  | 0 |
  TC 5, Week 32, n=0, 5, 0 |  | 0 |
  TC 5, Week 40, n=0, 1, 0 |  | 0 |
  TC 6, Week 8, n=0, 6, 0 |  | 0 |
  TC 6, Week 16, n=0, 6, 0 |  | 0 |
  TC 6, Week 24, n=0, 5, 0 |  | 0 |
  TC 6, Week 32, n=0, 3, 0 |  | 0 |

36. Secondary Outcome: Number of Participants With a CD3+ Cell Count Greater Than or Equal to the Lower Limit of Normal or the Baseline Value at the Indicated Time Point, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The number of participants with a CD3+ cell count greater than or equal to the lower limit of normal (LLN; reference range 0.11 to 0.66 gill per liter) or the baseline value (whichever was lower) is presented. The baseline assessment is defined as the start of the Double-blind Period.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 136 | 0
Participants
  TC 1, Week 8, n=0, 136, 0 |  | 115 |
  TC 1, Week 16, n=0, 100, 0 |  | 79 |
  TC 1, Week 24, n=0, 99, 0 |  | 75 |
  TC 1, Week 32, n=0, 50, 0 |  | 44 |
  TC 1, Week 40, n=0, 30, 0 |  | 27 |
  TC 1, Week 48, n=0, 23, 0 |  | 21 |
  TC 1, Week 56, n=0, 14, 0 |  | 11 |
  TC 1, Week 64, n=0, 7, 0 |  | 7 |
  TC 1, Week 72, n=0, 4, 0 |  | 4 |
  TC 1, Week 80, n=0, 1, 0 |  | 1 |
  TC 1, Week 88, n=0, 1, 0 |  | 1 |
  TC 1, Week 96, n=0, 1, 0 |  | 1 |
  TC 1, Week 104, n=0, 2, 0 |  | 2 |
  TC 1, Week 112, n=0, 1, 0 |  | 1 |
  TC 1, Week 120, n=0, 1, 0 |  | 1 |
  TC 1, Week 128, n=0, 1, 0 |  | 1 |
  TC 1, Week 144, n=0, 1, 0 |  | 1 |
  TC 2, Week 8, n=0, 93, 0 |  | 78 |
  TC 2, Week 16, n=0, 80, 0 |  | 70 |
  TC 2, Week 24, n=0, 70, 0 |  | 58 |
  TC 2, Week 32, n=0, 31, 0 |  | 29 |
  TC 2, Week 40, n=0, 20, 0 |  | 16 |
  TC 2, Week 48, n=0, 11, 0 |  | 9 |
  TC 2, Week 56, n=0, 8, 0 |  | 7 |
  TC 2, Week 64, n=0, 6, 0 |  | 4 |
  TC 2, Week 72, n=0, 2, 0 |  | 2 |
  TC 2, Week 80, n=0, 2, 0 |  | 2 |
  TC 2, Week 96, n=0, 1, 0 |  | 1 |
  TC 3, Week 8, n=0, 60, 0 |  | 49 |
  TC 3, Week 16, n=0, 45, 0 |  | 36 |
  TC 3, Week 24, n=0, 29, 0 |  | 22 |
  TC 3, Week 32, n=0, 12, 0 |  | 10 |
  TC 3, Week 40, n=0, 4, 0 |  | 2 |
  TC 3, Week 48, n=0, 2, 0 |  | 1 |
  TC 3, Week 56, n=0, 1, 0 |  | 1 |
  TC 4, Week 8, n=0, 29, 0 |  | 24 |
  TC 4, Week 16, n=0, 24, 0 |  | 20 |
  TC 4, Week 24, n=0, 13, 0 |  | 11 |
  TC 4, Week 32, n=0, 4, 0 |  | 3 |
  TC 4, Week 40, n=0, 1, 0 |  | 1 |
  TC 4, Week 48, n=0, 1, 0 |  | 1 |
  TC 5, Week 8, n=0, 13, 0 |  | 10 |
  TC 5, Week 16, n=0, 8, 0 |  | 7 |
  TC 5, Week 24, n=0, 5, 0 |  | 4 |
  TC 5, Week 32, n=0, 5, 0 |  | 4 |
  TC 5, Week 40, n=0, 1, 0 |  | 1 |
  TC 6, Week 8, n=0, 6, 0 |  | 5 |
  TC 6, Week 16, n=0, 6, 0 |  | 5 |
  TC 6, Week 24, n=0, 5, 0 |  | 5 |
  TC 6, Week 32, n=0, 3, 0 |  | 3 |

37. Secondary Outcome: Number of Participants With a CD4+ Cell Count Greater Than or Equal to the Lower Limit of Normal or the Baseline Value at the Indicated Time Point , During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The number of participants with a CD4+ cell count greater than or equal to the lower limit of normal (LLN; reference range 0.11 to 0.66 gill per liter) or the baseline value (whichever was lower) is presented. The baseline assessment is defined as the start of the Double-blind Period.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 136 | 0
Participants
  TC 1, Week 8, n=0, 136, 0 |  | 118 |
  TC 1, Week 16, n=0, 100, 0 |  | 83 |
  TC 1, Week 24, n=0, 99, 0 |  | 80 |
  TC 1, Week 32, n=0, 50, 0 |  | 45 |
  TC 1, Week 40, n=0, 30, 0 |  | 27 |
  TC 1, Week 48, n=0, 23, 0 |  | 21 |
  TC 1, Week 56, n=0, 14, 0 |  | 13 |
  TC 1, Week 64, n=0, 7, 0 |  | 7 |
  TC 1, Week 72, n=0, 4, 0 |  | 4 |
  TC 1, Week 80, n=0, 1, 0 |  | 1 |
  TC 1, Week 88, n=0, 1, 0 |  | 1 |
  TC 1, Week 96, n=0, 1, 0 |  | 1 |
  TC 1, Week 104, n=0, 2, 0 |  | 2 |
  TC 1, Week 112, n=0, 1, 0 |  | 1 |
  TC 1, Week 120, n=0, 1, 0 |  | 1 |
  TC 1, Week 128, n=0, 1, 0 |  | 1 |
  TC 1, Week 144, n=0, 1, 0 |  | 1 |
  TC 2, Week 8, n=0, 93, 0 |  | 81 |
  TC 2, Week 16, n=0, 80, 0 |  | 67 |
  TC 2, Week 24, n=0, 70, 0 |  | 62 |
  TC 2, Week 32, n=0, 31, 0 |  | 29 |
  TC 2, Week 40, n=0, 20, 0 |  | 16 |
  TC 2, Week 48, n=0, 11, 0 |  | 9 |
  TC 2, Week 56, n=0, 8, 0 |  | 7 |
  TC 2, Week 64, n=0, 6, 0 |  | 4 |
  TC 2, Week 72, n=0, 2, 0 |  | 2 |
  TC 2, Week 80, n=0, 2, 0 |  | 2 |
  TC 2, Week 96, n=0, 1, 0 |  | 1 |
  TC 3, Week 8, n=0, 60, 0 |  | 49 |
  TC 3, Week 16, n=0, 45, 0 |  | 36 |
  TC 3, Week 24, n=0, 29, 0 |  | 23 |
  TC 3, Week 32, n=0, 12, 0 |  | 11 |
  TC 3, Week 40, n=0, 4, 0 |  | 3 |
  TC 3, Week 48, n=0, 2, 0 |  | 2 |
  TC 3, Week 56, n=0, 1, 0 |  | 1 |
  TC 4, Week 8, n=0, 29, 0 |  | 26 |
  TC 4, Week 16, n=0, 24, 0 |  | 20 |
  TC 4, Week 24, n=0, 13, 0 |  | 11 |
  TC 4, Week 32, n=0, 4, 0 |  | 3 |
  TC 4, Week 40, n=0, 1, 0 |  | 1 |
  TC 4, Week 48, n=0, 1 |  | 1 |
  TC 5, Week 8, n=0, 13, 0 |  | 12 |
  TC 5, Week 16, n=0, 8, 0 |  | 8 |
  TC 5, Week 24, n=0, 5, 0 |  | 5 |
  TC 5, Week 32, n=0, 5, 0 |  | 5 |
  TC 5, Week 40, n=0, 1, 0 |  | 1 |
  TC 6, Week 8, n=0, 6, 0 |  | 5 |
  TC 6, Week 16, n=0, 6, 0 |  | 6 |
  TC 6, Week 24, n=0, 5, 0 |  | 5 |
  TC 6, Week 32, n=0, 3, 0 |  | 3 |

38. Secondary Outcome: Number of Participants With a CD8+ Cell Count Greater Than or Equal to the Lower Limit of Normal or the Baseline Value at the Indicated Time Point , During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The number of participants with a CD8+ cell count greater than or equal to the lower limit of normal (LLN; reference range 0.11 to 0.66 gill per liter) or the baseline value (whichever was lower) is presented. The baseline assessment is defined as the start of the Double-blind Period.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 136 | 0
Participants
  TC 1, Week 8, n=0, 136, 0 |  | 121 |
  TC 1, Week 16, n=0, 100, 0 |  | 86 |
  TC 1, Week 24, n=0, 99, 0 |  | 87 |
  TC 1, Week 32, n=0, 50, 0 |  | 47 |
  TC 1, Week 40, n=0, 30, 0 |  | 27 |
  TC 1, Week 48, n=0, 23, 0 |  | 20 |
  TC 1, Week 56, n=0, 14, 0 |  | 13 |
  TC 1, Week 64, n=0, 7, 0 |  | 7 |
  TC 1, Week 72, n=0, 4, 0 |  | 4 |
  TC 1, Week 80, n=0, 1, 0 |  | 1 |
  TC 1, Week 88, n=0, 1, 0 |  | 1 |
  TC 1, Week 96, n=0, 1, 0 |  | 1 |
  TC 1, Week 104, n=0, 2, 0 |  | 2 |
  TC 1, Week 112, n=0, 1, 0 |  | 1 |
  TC 1, Week 120, n=0, 1, 0 |  | 1 |
  TC 1, Week 128, n=0, 1, 0 |  | 1 |
  TC 1, Week 144, n=0, 1, 0 |  | 1 |
  TC 2, Week 8, n=0, 93, 0 |  | 82 |
  TC 2, Week 16, n=0, 80, 0 |  | 74 |
  TC 2, Week 24, n=0, 70, 0 |  | 63 |
  TC 2, Week 32, n=0, 31, 0 |  | 29 |
  TC 2, Week 40, n=0, 20, 0 |  | 19 |
  TC 2, Week 48, n=0, 11, 0 |  | 11 |
  TC 2, Week 56, n=0, 8, 0 |  | 7 |
  TC 2, Week 64, n=0, 6, 0 |  | 5 |
  TC 2, Week 72, n=0, 2, 0 |  | 2 |
  TC 2, Week 80, n=0, 2, 0 |  | 2 |
  TC 2, Week 96, n=0, 1, 0 |  | 1 |
  TC 3, Week 8, n=0, 60, 0 |  | 54 |
  TC 3, Week 16, n=0, 45, 0 |  | 43 |
  TC 3, Week 24, n=0, 29, 0 |  | 24 |
  TC 3, Week 32, n=0, 12, 0 |  | 12 |
  TC 3, Week 40, n=0, 4, 0 |  | 3 |
  TC 3, Week 48, n=0, 2, 0 |  | 1 |
  TC 3, Week 56, n=0, 1, 0 |  | 1 |
  TC 4, Week 8, n=0, 29, 0 |  | 26 |
  TC 4, Week 16, n=0, 24, 0 |  | 23 |
  TC 4, Week 24, n=0, 13, 0 |  | 13 |
  TC 4, Week 32, n=0, 4, 0 |  | 4 |
  TC 4, Week 40, n=0, 1, 0 |  | 1 |
  TC 4, Week 48, n=0, 1, 0 |  | 1 |
  TC 5, Week 8, n=0, 13, 0 |  | 13 |
  TC 5, Week 16, n=0, 8, 0 |  | 8 |
  TC 5, Week 24, n=0, 5, 0 |  | 5 |
  TC 5, Week 32, n=0, 5, 0 |  | 5 |
  TC 5, Week 40, n=0, 1, 0 |  | 1 |
  TC 6, Week 8, n=0, 6, 0 |  | 5 |
  TC 6, Week 16, n=0, 6, 0 |  | 5 |
  TC 6, Week 24, n=0, 5, 0 |  | 5 |
  TC 6, Week 32, n=0, 3, 0 |  | 2 |

39. Secondary Outcome: Number of Participants With the Indicated Clinical Chemistry Values of Potential Clinical Concern at Baseline or Any Visit Post-baseline, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: Only those parameters for which at least one value of clinical concern (CC) was reported are summarized. The baseline (BL) value for a treatment course is defined as the latest value on or before the date of infusion A of the treatment course. The post-baseline (PBL) visit is defined as any visit after the date of infusion A during the specified treatment course. Pre-defined limits of potential clinical concern (CC Low [relative to the lower limit of normal], CC High [relative to the upper limit of normal]) are: Albumin: 0.9, 1.5; Alanine amino transferase (ALT): NA, 2; Alkaline phosphatase (ALP): NA, 1.5; Aspartate amino transferase (AST): NA, 2; Bilirubin total (TBIL): NA, 1.5; Calcium: 0.85, 1.08; CO2 content/bicarbonate (BCO): 0.85, 1.2; Creatine kinase (CK): NA, 2; Creatinine: NA, 1.2; Gamma glutamyl transferase (GGT): NA, 2; Potassium: 0.9, 1.1; Urea/blood urea nitrogen (BUN): NA, 1.5; Uric acid: NA, 1.5.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 144 | 0
Participants
  Albumin, TC 1, BL, CC low, n=0, 144, 0 |  | 1 |
  Albumin, TC 1, PBL, CC low, n=0, 136, 0 |  | 1 |
  ALT, TC 1, BL, CC high, n=0, 144, 0 |  | 1 |
  ALT, TC 1, PBL, CC high, n=0, 136, 0 |  | 6 |
  ALP, TC 1, BL, CC high, n=0, 144, 0 |  | 0 |
  ALP, TC 1, PBL, CC high, n=0, 136, 0 |  | 4 |
  AST, TC 1, BL, CC high, n=0, 142, 0 |  | 0 |
  AST, TC 1, PBL, CC high, n=0, 136, 0 |  | 2 |
  TBIL, TC 1, BL, CC high, n=0, 144, 0 |  | 0 |
  TBIL, TC 1, PBL, CC high, n=0, 136, 0 |  | 0 |
  Calcium, TC 1, BL, CC low, n=0, 142, 0 |  | 0 |
  Calcium, TC 1, PBL, CC low, n=0, 136, 0 |  | 2 |
  Calcium, TC 1, BL, CC high, n=0, 142, 0 |  | 0 |
  Calcium, TC 1, PBL, CC high, n=0, 136, 0 |  | 0 |
  CO2/BCO, TC 1, BL, CC low, n=0, 142, 0 |  | 5 |
  CO2/BCO, TC 1, PBL, CC low, n=0, 136, 0 |  | 9 |
  CK, TC 1, BL, CC high, n=0, 144, 0 |  | 0 |
  CK, TC 1, PBL, CC high, n=0, 136, 0 |  | 1 |
  Creatinine, TC 1, BL, CC high, n=0, 144, 0 |  | 0 |
  Creatinine, TC 1,PBL, CC high, n=0, 136, 0 |  | 1 |
  GGT, TC 1, BL, CC high, n=0, 144, 0 |  | 7 |
  GGT, TC 1, PBL, CC high, n=0, 136, 0 |  | 8 |
  Potassium, TC 1, BL, CC high, n=0, 142, 0 |  | 2 |
  Potassium, TC 1, PBL, CC high, n=0, 136, 0 |  | 0 |
  Potassium, TC 1, BL, CC low, n=0, 142, 0 |  | 1 |
  Potassium, TC 1, PBL, CC low, n=0, 136, 0 |  | 1 |
  Urea/BUN, TC 1, BL, CC high, n=0, 144, 0 |  | 2 |
  Urea/BUN, TC 1, PBL, CC high, n=0, 136, 0 |  | 3 |
  Uric acid, TC 1, BL, CC high, n=0, 144, 0 |  | 0 |
  Uric acid, TC 1, PBL, CC high, n=0, 136, 0 |  | 0 |
  Albumin, TC 2, BL, CC low, n=0, 85, 0 |  | 0 |
  Albumin, TC 2, PBL, CC low, n=0, 92, 0 |  | 0 |
  ALT, TC 2, BL, CC high, n=0, 85, 0 |  | 1 |
  ALT, TC 2, PBL, CC high, n=0, 92, 0 |  | 5 |
  ALP, TC 2, BL, CC high, n=0, 85, 0 |  | 0 |
  ALP, TC 2, PBL, CC high, n=0, 92, 0 |  | 1 |
  AST, TC 2, BL, CC high, n=0, 85, 0 |  | 1 |
  AST, TC 2, PBL, CC high, n=0, 92, 0 |  | 2 |
  TBIL, TC 2, BL, CC high, n=0, 85, 0 |  | 0 |
  TBIL, TC 2, PBL, CC high, n=0, 92, 0 |  | 0 |
  Calcium, TC 2, BL, CC low, n=0, 85, 0 |  | 0 |
  Calcium, TC 2, PBL, CC low, n=0, 92, 0 |  | 0 |
  Calcium, TC 2, BL, CC high, n=0, 85, 0 |  | 0 |
  Calcium, TC 2, PBL, CC high, n=0, 92, 0 |  | 1 |
  CO2/BCO, TC 2, BL, CC low, n=0, 85, 0 |  | 1 |
  CO2/BCO, TC 2, PBL, CC low, n=0, 92 |  | 7 |
  CK, TC 2, BL, CC high, n=0, 85, 0 |  | 0 |
  CK, TC 2, PBL, CC high, n=0, 92, 0 |  | 0 |
  Creatinine, TC 2, BL, CC high, n=0, 85, 0 |  | 0 |
  Creatinine, TC 2,PBL, CC high, n=0, 92, 0 |  | 0 |
  GGT, TC 2, BL, CC high, n=0, 85, 0 |  | 3 |
  GGT, TC 2, PBL, CC high, n=0, 92, 0 |  | 3 |
  Potassium, TC 2, BL, CC high, n=0, 85, 0 |  | 1 |
  Potassium, TC 2, PBL, CC high, n=0, 92, 0 |  | 0 |
  Potassium, TC 2, BL, CC low, n=0, 85, 0 |  | 0 |
  Potassium, TC 2, PBL, CC low, n=0, 92, 0 |  | 0 |
  Urea/BUN, TC 2, BL, CC high, n=0, 85, 0 |  | 1 |
  Urea/BUN, TC 2, PBL, CC high, n=0, 92, 0 |  | 3 |
  Uric acid, TC 2, BL, CC high, n=0, 85, 0 |  | 0 |
  Uric acid, TC 2, PBL, CC high, n=0, 92, 0 |  | 1 |
  Albumin, TC 3, BL, CC low, n=0, 57, 0 |  | 0 |
  Albumin, TC 3, PBL, CC low, n=0, 62, 0 |  | 1 |
  ALT, TC 3, BL, CC high, n=0, 57, 0 |  | 1 |
  ALT, TC 3, PBL, CC high, n=0, 62, 0 |  | 1 |
  ALP, TC 3, BL, CC high, n=0, 57, 0 |  | 0 |
  ALP, TC 3, PBL, CC high, n=0, 62, 0 |  | 1 |
  AST, TC 3, BL, CC high, n=0, 57, 0 |  | 1 |
  AST, TC 3, PBL, CC high, n=0, 62, 0 |  | 0 |
  TBIL, TC 3, BL, CC high, n=0, 57, 0 |  | 0 |
  TBIL, TC 3, PBL, CC high, n=0, 62, 0 |  | 0 |
  Calcium, TC 3, BL, CC low, n=0, 57, 0 |  | 0 |
  Calcium, TC 3, PBL, CC low, n=0, 62, 0 |  | 0 |
  Calcium, TC 3, BL, CC high, n=0, 57, 0 |  | 1 |
  Calcium, TC 3, PBL, CC high, n=0, 62, 0 |  | 1 |
  CO2/BCO, TC 3, BL, CC low, n=0, 57, 0 |  | 0 |
  CO2/BCO, TC 3, PBL, CC low, n=0, 62, 0 |  | 2 |
  CK, TC 3, BL, CC high, n=0, 57, 0 |  | 0 |
  CK, TC 3, PBL, CC high, n=0, 62, 0 |  | 0 |
  Creatinine, TC 3, BL, CC high, n=0, 57, 0 |  | 0 |
  Creatinine, TC 3,PBL, CC high, n=0, 62, 0 |  | 0 |
  GGT, TC 3, BL, CC high, n=0, 57, 0 |  | 0 |
  GGT, TC 3, PBL, CC high, n=0, 62, 0 |  | 3 |
  Potassium, TC 3, BL, CC high, n=0, 57, 0 |  | 0 |
  Potassium, TC 3, PBL, CC high, n=0, 62, 0 |  | 0 |
  Potassium, TC 3, BL, CC low, n=0, 57, 0 |  | 0 |
  Potassium, TC 3, PBL, CC low, n=0, 62, 0 |  | 0 |
  Urea/BUN, TC 3, BL, CC high, n=0, 57, 0 |  | 0 |
  Urea/BUN, TC 3, PBL, CC high, n=0, 62, 0 |  | 0 |
  Uric acid, TC 3, BL, CC high, n=0, 57, 0 |  | 0 |
  Uric acid, TC 3, PBL, CC high, n=0, 62, 0 |  | 0 |
  Albumin, TC 4, BL, CC low, n=0, 28, 0 |  | 0 |
  Albumin, TC 4, PBL, CC low, n=0, 29, 0 |  | 0 |
  ALT, TC 4, BL, CC high, n=0, 28, 0 |  | 0 |
  ALT, TC 4, PBL, CC high, n=0, 29, 0 |  | 0 |
  ALP, TC 4, BL, CC high, n=0, 28, 0 |  | 1 |
  ALP, TC 4, PBL, CC high, n=0, 29, 0 |  | 1 |
  AST, TC 4, BL, CC high, n=0, 28, 0 |  | 0 |
  AST, TC 4, PBL, CC high, n=0, 29, 0 |  | 0 |
  TBIL, TC 4, BL, CC high, n=0, 28, 0 |  | 0 |
  TBIL, TC 4, PBL, CC high, n=0, 29, 0 |  | 1 |
  Calcium, TC 4, BL, CC low, n=0, 28, 0 |  | 0 |
  Calcium, TC 4, PBL, CC low, n=0, 29, 0 |  | 0 |
  Calcium, TC 4, BL, CC high, n=0, 28, 0 |  | 0 |
  Calcium, TC 4, PBL, CC high, n=0, 29, 0 |  | 0 |
  CO2/BCO, TC 4, BL, CC low, n=0, 28, 0 |  | 1 |
  CO2/BCO, TC 4, PBL, CC low, n=0, 29, 0 |  | 1 |
  CK, TC 4, BL, CC high, n=0, 28, 0 |  | 0 |
  CK, TC 4, PBL, CC high, n=0, 29, 0 |  | 0 |
  Creatinine, TC 4, BL, CC high, n=0, 28, 0 |  | 0 |
  Creatinine, TC 4,PBL, CC high, n=0, 29, 0 |  | 0 |
  GGT, TC 4, BL, CC high, n=0, 28, 0 |  | 2 |
  GGT, TC 4, PBL, CC high, n=0, 29, 0 |  | 1 |
  Potassium, TC 4, BL, CC high, n=0, 28, 0 |  | 0 |
  Potassium, TC 4, PBL, CC high, n=0, 29, 0 |  | 0 |
  Potassium, TC 4, BL, CC low, n=0, 28, 0 |  | 0 |
  Potassium, TC 4, PBL, CC low, n=0, 29, 0 |  | 0 |
  Urea/BUN, TC 4, BL, CC high, n=0, 28, 0 |  | 0 |
  Urea/BUN, TC 4, PBL, CC high, n=0, 29, 0 |  | 0 |
  Uric acid, TC 4, BL, CC high, n=0, 28, 0 |  | 0 |
  Uric acid, TC 4, PBL, CC high, n=0, 29, 0 |  | 0 |
  Albumin, TC 5, BL, CC low, n=0, 12, 0 |  | 0 |
  Albumin, TC 5, PBL, CC low, n=0, 13, 0 |  | 0 |
  ALT, TC 5, BL, CC high, n=0, 12 |  | 0 |
  ALT, TC 5, PBL, CC high, n=0, 13, 0 |  | 0 |
  ALP, TC 5, BL, CC high, n=0, 12, 0 |  | 0 |
  ALP, TC 5, PBL, CC high, n=0, 13, 0 |  | 0 |
  AST, TC 5, BL, CC high, n=0, 12, 0 |  | 0 |
  AST, TC 5, PBL, CC high, n=0, 13, 0 |  | 0 |
  TBIL, TC 5, BL, CC high, n=0, 12, 0 |  | 0 |
  TBIL, TC 5, PBL, CC high, n=0, 13, 0 |  | 1 |
  Calcium, TC 5, BL, CC low, n=0, 12, 0 |  | 0 |
  Calcium, TC 5, PBL, CC low, n=0, 13, 0 |  | 0 |
  Calcium, TC 5, BL, CC high, n=0, 12, 0 |  | 0 |
  Calcium, TC 5, PBL, CC high, n=0, 13, 0 |  | 0 |
  CO2/BCO, TC 5, BL, CC low, n=0, 12, 0 |  | 0 |
  CO2/BCO, TC 5, PBL, CC low, n=0, 13, 0 |  | 1 |
  CK, TC 5, BL, CC high, n=0, 12, 0 |  | 0 |
  CK, TC 5, PBL, CC high, n=0, 13, 0 |  | 0 |
  Creatinine, TC 5, BL, CC high, n=0, 12, 0 |  | 0 |
  Creatinine, TC 5,PBL, CC high, n=0, 13, 0 |  | 0 |
  GGT, TC 5, BL, CC high, n=0, 12, 0 |  | 1 |
  GGT, TC 5, PBL, CC high, n=0, 13, 0 |  | 1 |
  Potassium, TC 5, BL, CC high, n=0, 12, 0 |  | 0 |
  Potassium, TC 5, PBL, CC high, n=0, 13, 0 |  | 0 |
  Potassium, TC 5, BL, CC low, n=0, 12, 0 |  | 0 |
  Potassium, TC 5, PBL, CC low, n=0, 13, 0 |  | 0 |
  Urea/BUN, TC 5, BL, CC high, n=0, 12, 0 |  | 0 |
  Urea/BUN, TC 5, PBL, CC high, n=0, 13, 0 |  | 0 |
  Uric acid, TC 5, BL, CC high, n=0, 12, 0 |  | 0 |
  Uric acid, TC 5, PBL, CC high, n=0, 13, 0 |  | 0 |
  Albumin, TC 6, BL, CC low, n=0, 6, 0 |  | 0 |
  Albumin, TC 6, PBL, CC low, n=0, 6, 0 |  | 0 |
  ALT, TC 6, BL, CC high, n=0, 6, 0 |  | 0 |
  ALT, TC 6, PBL, CC high, n=0, 6, 0 |  | 0 |
  ALP, TC 6, BL, CC high, n=0, 6, 0 |  | 0 |
  ALP, TC 6, PBL, CC high, n=0, 6, 0 |  | 1 |
  AST, TC 6, BL, CC high, n=0, 6, 0 |  | 0 |
  AST, TC 6, PBL, CC high, n=0, 6, 0 |  | 0 |
  TBIL, TC 6, BL, CC high, n=0, 6, 0 |  | 1 |
  TBIL, TC 6, PBL, CC high, n=0, 6, 0 |  | 0 |
  Calcium, TC 6, BL, CC low, n=0, 6, 0 |  | 0 |
  Calcium, TC 6, PBL, CC low, n=0, 6, 0 |  | 0 |
  Calcium, TC 6, BL, CC high, n=0, 6, 0 |  | 0 |
  Calcium, TC 6, PBL, CC high, n=0, 6, 0 |  | 0 |
  CO2/BCO, TC 6, BL, CC low, n=0, 6, 0 |  | 0 |
  CO2/BCO, TC 6, PBL, CC low, n=0, 6, 0 |  | 0 |
  CK, TC 6, BL, CC high, n=0, 6, 0 |  | 0 |
  CK, TC 6, PBL, CC high, n=0, 6, 0 |  | 0 |
  Creatinine, TC , BL, CC high, n=0, 6, 0 |  | 0 |
  Creatinine, TC 6,PBL, CC high, n=0, 6, 0 |  | 0 |
  GGT, TC 6, BL, CC high, n=0, 6, 0 |  | 0 |
  GGT, TC 6, PBL, CC high, n=0, 6, 0 |  | 0 |
  Potassium, TC 6, BL, CC high, n=0, 6, 0 |  | 0 |
  Potassium, TC 6, PBL, CC high, n=0, 6, 0 |  | 0 |
  Potassium, TC 6, BL, CC low, n=0, 6, 0 |  | 0 |
  Potassium, TC 6, PBL, CC low, n=0, 6, 0 |  | 0 |
  Urea/BUN, TC 6, BL, CC high, n=0, 6, 0 |  | 0 |
  Urea/BUN, TC 6, PBL, CC high, n=0, 6, 0 |  | 0 |
  Uric acid, TC 6, BL, CC high, n=0, 6, 0 |  | 0 |
  Uric acid, TC 6, PBL, CC high, n=0, 6, 0 |  | 0 |

40. Secondary Outcome: Number of Participants With the Indicated Hematology Values of Potential Clinical Concern at Baseline or Any Visit Post-baseline, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: Only those parameters for which at least one value of clinical concern (CC) was reported are summarized. The baseline (BL) value for a treatment course is defined as the latest value on or before the date of infusion A of the treatment course. The post-baseline (PBL) visit is defined as any visit after the date of infusion A during the specified treatment course. Pre-defined limits of potential clinical concern (CC Low [relative to lower limit of normal], CC High [relative to upper limit of normal]) are: Eosinophils: NA, 2; Hematocrit (HCT): 0.75, 1.2; Hemoglobin (Hb): 0.75, 1.2; Monocytes: 0.2, 5 2; Neutrophils total (TNUE): 0.8, 1.6; Platelet count (PC): 0.65, 1.5; Red blood cell count (RBC): 0.7, 5 2; White blood cell count (WBC): 0.7, 1.6.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 143 | 0
Participants
  Eosinophils, TC 1, BL,CC high, n=0, 143, 0 |  | 1 |
  Eosinophils, TC 1,PBL,CC high, n=0, 136, 0 |  | 1 |
  HCT, TC 1, BL, CC low, n=0, 143, 0 |  | 0 |
  HCT, TC 1, PBL, CC low, n=0, 136, 0 |  | 1 |
  Hb, TC 1, BL, CC low, n=0, 143, 0 |  | 1 |
  Hb, TC 1, PBL, CC low, n=0, 136, 0 |  | 5 |
  Monocytes, TC 1, BL, CC low, n=0, 143, 0 |  | 2 |
  Monocytes, TC 1, PBL, CC low, n=0, 136, 0 |  | 13 |
  Monocytes, TC 1, BL, CC high, n=0, 143, 0 |  | 0 |
  Monocytes, TC 1, PBL, CC high, n=0, 136, 0 |  | 0 |
  PC, TC 1, BL, CC low, n=0, 141, 0 |  | 0 |
  PC, TC 1, PBL, CC low, n=0, 136, 0 |  | 0 |
  PC, TC 1, BL, CC high, n=0, 141, 0 |  | 0 |
  PC, TC 1, PBL, CC high, n=0, 136, 0 |  | 1 |
  RBC count, TC 1, BL, CC low, n=0, 143, 0 |  | 1 |
  RBC count, TC 1, PBL, CC low, n=0, 136, 0 |  | 2 |
  TNUE, TC 1, BL, CC low, n=0, 142, 0 |  | 0 |
  TNUE, TC 1, PBL, CC low, n=0, 136, 0 |  | 0 |
  TNUE, TC 1, BL, CC high, n=0, 142, 0 |  | 0 |
  TNUE, TC 1,PBL, CC high, n=0, 136, 0 |  | 3 |
  WBC count, TC 1, BL, CC low, n=0, 143, 0 |  | 0 |
  WBC count, TC 1, PBL, CC low, n=0, 136, 0 |  | 0 |
  WBC count, TC 1, BL, CC high, n=0, 143, 0 |  | 0 |
  WBC count, TC 1, PBL, CC high, n=0, 136, 0 |  | 1 |
  Eosinophils, TC 2, BL,CC high, n=0, 85, 0 |  | 0 |
  Eosinophils, TC 2,PBL,CC high, n=0, 93, 0 |  | 0 |
  HCT, TC 2, BL, CC low, n=0, 85, 0 |  | 0 |
  HCT, TC 2, PBL, CC low, n=0, 93, 0 |  | 0 |
  Hb, TC 2, BL, CC low, n=0, 85, 0 |  | 1 |
  Hb, TC 2, PBL, CC low, n=0, 93, 0 |  | 1 |
  Monocytes, TC 2, BL, CC low, n=0, 85, 0 |  | 2 |
  Monocytes, TC 2, PBL, CC low, n=0, 93, 0 |  | 1 |
  Monocytes, TC 2, BL, CC high, n=0, 85, 0 |  | 0 |
  Monocytes, TC 2, PBL, CC high, n=0, 93, 0 |  | 1 |
  PC, TC 2, BL, CC low, n=0, 84, 0 |  | 0 |
  PC, TC 2, PBL, CC low, n=0, 93, 0 |  | 1 |
  PC, TC 2, BL, CC high, n=0, 84, 0 |  | 0 |
  PC, TC 2, PBL, CC high, n=0, 93, 0 |  | 0 |
  RBC count, TC 2, BL, CC low, n=0, 85, 0 |  | 1 |
  RBC count, TC 2, PBL, CC low, n=0, 93, 0 |  | 1 |
  TNUE, TC 2, BL, CC low, n=0, 85, 0 |  | 0 |
  TNUE, TC 2, PBL, CC low, n=0, 92, 0 |  | 1 |
  TNUE, TC 2, BL, CC high, n=0, 85, 0 |  | 1 |
  TNUE, TC 2,PBL, CC high, n=0, 92, 0 |  | 0 |
  WBC count, TC 2, BL, CC low, n=0, 85, 0 |  | 0 |
  WBC count, TC 2, PBL, CC low, n=0, 93, 0 |  | 1 |
  WBC count, TC 2, BL, CC high, n=0, 85, 0 |  | 1 |
  WBC count, TC 2, PBL, CC high, n=0, 93, 0 |  | 0 |
  Eosinophils, TC 3, BL,CC high, n=0, 58, 0 |  | 0 |
  Eosinophils, TC 3,PBL,CC high, n=0, 62, 0 |  | 0 |
  HCT, TC 3, BL, CC low, n=0, 58, 0 |  | 0 |
  HCT, TC 3, PBL, CC low, n=0, 62, 0 |  | 0 |
  Hb, TC 3, BL, CC low, n=0, 58, 0 |  | 0 |
  Hb, TC 3, PBL, CC low, n=0, 62, 0 |  | 1 |
  Monocytes, TC 3, BL, CC low, n=0, 58, 0 |  | 1 |
  Monocytes, TC 3, PBL, CC low, n=0, 62, 0 |  | 3 |
  Monocytes, TC 3, BL, CC high, n=0, 58, 0 |  | 0 |
  Monocytes, TC 3, PBL, CC high, n=0, 62, 0 |  | 0 |
  PC, TC 3, BL, CC low, n=0, 57, 0 |  | 1 |
  PC, TC 3, PBL, CC low, n=0, 62, 0 |  | 1 |
  PC, TC 3, BL, CC high, n=0, 57, 0 |  | 0 |
  PC, TC 3, PBL, CC high, n=0, 62, 0 |  | 0 |
  RBC count, TC 3, BL, CC low, n=0, 58, 0 |  | 0 |
  RBC count, TC 3, PBL, CC low, n=0, 62, 0 |  | 0 |
  TNUE, TC 3, BL, CC low, n=0, 57, 0 |  | 0 |
  TNUE, TC 3, PBL, CC low, n=0, 60, 0 |  | 0 |
  TNUE, TC 3, BL, CC high, n=0, 57, 0 |  | 0 |
  TNUE, TC 3,PBL, CC high, n=0, 60, 0 |  | 0 |
  WBC count, TC 3, BL, CC low, n=0, 58, 0 |  | 0 |
  WBC count, TC 3, PBL, CC low, n=0, 62, 0 |  | 0 |
  WBC count, TC 3, BL, CC high, n=0, 58, 0 |  | 0 |
  WBC count, TC 4, PBL, CC high, n=0, 62, 0 |  | 0 |
  Eosinophils, TC 4, BL,CC high, n=0, 28, 0 |  | 0 |
  Eosinophils, TC 4,PBL,CC high, n=0, 29, 0 |  | 0 |
  HCT, TC 4, BL, CC low, n=0, 28, 0 |  | 0 |
  HCT, TC 4, PBL, CC low, n=0, 29, 0 |  | 0 |
  Hb, TC 4, BL, CC low, n=0, 28, 0 |  | 1 |
  Hb, TC 1, PBL, CC low, n=0, 29, 0 |  | 0 |
  Monocytes, TC 4, BL, CC low, n=0, 28, 0 |  | 1 |
  Monocytes, TC 4, PBL, CC low, n=0, 29, 0 |  | 0 |
  Monocytes, TC 4, BL, CC high, n=0, 28, 0 |  | 0 |
  Monocytes, TC 4, PBL, CC high, n=0, 29, 0 |  | 0 |
  PC, TC 4, BL, CC low, n=0, 28, 0 |  | 0 |
  PC, TC 4, PBL, CC low, n=0, 29, 0 |  | 0 |
  PC, TC 4, BL, CC high, n=0, 28, 0 |  | 0 |
  PC, TC 4, PBL, CC high, n=0, 29, 0 |  | 0 |
  RBC count, TC 4, BL, CC low, n=0, 28, 0 |  | 1 |
  RBC count, TC 4, PBL, CC low, n=0, 29, 0 |  | 0 |
  TNUE, TC 4, BL, CC low, n=0, 26, 0 |  | 0 |
  TNUE, TC 4, PBL, CC low, n=0, 28, 0 |  | 0 |
  TNUE, TC 4, BL, CC high, n=0, 26, 0 |  | 0 |
  TNUE, TC 4,PBL, CC high, n=0, 28, 0 |  | 0 |
  WBC count, TC 4, BL, CC low, n=0, 28, 0 |  | 0 |
  WBC count, TC 4, PBL, CC low, n=0, 29, 0 |  | 0 |
  WBC count, TC 4, BL, CC high, n=0, 28, 0 |  | 0 |
  WBC count, TC 4, PBL, CC high, n=0, 29, 0 |  | 0 |
  Eosinophils, TC 5, BL,CC high, n=0, 12, 0 |  | 0 |
  Eosinophils, TC 5,PBL,CC high, n=0, 13, 0 |  | 0 |
  HCT, TC 5, BL, CC low, n=0, 12, 0 |  | 0 |
  HCT, TC 5, PBL, CC low, n=0, 13, 0 |  | 0 |
  Hb, TC 5, BL, CC low, n=0, 12 |  | 0 |
  Hb, TC 5, PBL, CC low, n=0, 13, 0 |  | 0 |
  Monocytes, TC 5, BL, CC low, n=0, 12, 0 |  | 0 |
  Monocytes, TC 5, PBL, CC low, n=0, 13, 0 |  | 0 |
  Monocytes, TC 5, BL, CC high, n=0, 12, 0 |  | 0 |
  Monocytes, TC 5, PBL, CC high, n=0, 13, 0 |  | 0 |
  PC, TC 5, BL, CC low, n=0, 12, 0 |  | 0 |
  PC, TC 5, PBL, CC low, n=0, 13, 0 |  | 0 |
  PC, TC 5, BL, CC high, n=0, 12, 0 |  | 0 |
  PC, TC 5, PBL, CC high, n=0, 13, 0 |  | 0 |
  RBC count, TC 5, BL, CC low, n=0, 12, 0 |  | 0 |
  RBC count, TC 5, PBL, CC low, n=0, 13, 0 |  | 0 |
  TNUE, TC 5, BL, CC low, n=0, 11, 0 |  | 0 |
  TNUE, TC 5, PBL, CC low, n=0, 13 |  | 0 |
  TNUE, TC 5, BL, CC high, n=0, 11 |  | 0 |
  TNUE, TC 5,PBL, CC high, n=0, 13, 0 |  | 0 |
  WBC count, TC 5, BL, CC low, n=0, 12, 0 |  | 0 |
  WBC count, TC 5, PBL, CC low, n=0, 13, 0 |  | 0 |
  WBC count, TC 5, BL, CC high, n=0, 12, 0 |  | 0 |
  WBC count, TC 5, PBL, CC high, n=0, 13, 0 |  | 0 |
  Eosinophils, TC 6, BL,CC high, n=0, 6, 0 |  | 0 |
  Eosinophils, TC 6,PBL,CC high, n=0, 6, 0 |  | 0 |
  HCT, TC 6, BL, CC low, n=0, 6, 0 |  | 0 |
  HCT, TC 6, PBL, CC low, n=0, 6, 0 |  | 0 |
  Hb, TC 6, BL, CC low, n=0, 6, 0 |  | 0 |
  Hb, TC 6, PBL, CC low, n=0, 6, 0 |  | 0 |
  Monocytes, TC 6, BL, CC low, n=0, 6, 0 |  | 0 |
  Monocytes, TC 6, PBL, CC low, n=0, 6, 0 |  | 0 |
  Monocytes, TC 6, BL, CC high, n=0, 6, 0 |  | 0 |
  Monocytes, TC 6, PBL, CC high, n=0, 6, 0 |  | 0 |
  PC, TC 6, BL, CC low, n=0, 6, 0 |  | 0 |
  PC, TC 6, PBL, CC low, n=0, 6, 0 |  | 0 |
  PC, TC 6, BL, CC high, n=0, 6, 0 |  | 0 |
  PC, TC 6, PBL, CC high, n=0, 6, 0 |  | 0 |
  RBC count, TC 6, BL, CC low, n=0, 6, 0 |  | 0 |
  RBC count, TC 6, PBL, CC low, n=0, 6, 0 |  | 0 |
  TNUE, TC 6, BL, CC low, n=0, 6, 0 |  | 0 |
  TNUE, TC 6, PBL, CC low, n=0, 6, 0 |  | 0 |
  TNUE, TC 6, BL, CC high, n=0, 6, 0 |  | 0 |
  TNUE, TC 6,PBL, CC high, n=0, 6, 0 |  | 0 |
  WBC count, TC 6, BL, CC low, n=0, 6, 0 |  | 0 |
  WBC count, TC 6, PBL, CC low, n=0, 6, 0 |  | 0 |
  WBC count, TC 6, BL, CC high, n=0, 6, 0 |  | 0 |
  WBC count, TC 6, PBL, CC high, n=0, 6, 0 |  | 0 |

41. Secondary Outcome: Number of Participants With Vital Sign Data Outside the Clinical Concern Range at Baseline or Any Visit Post-baseline, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The baseline value for a treatment course is defined as the value before infusion A of each treatment course. The post-baseline visit is defined as any assessment during or after the start of infusion A during the specified treatment course. Pre-defined limits of potential clinical concern for vital signs (Low, High) are: Diastolic blood pressure (DBP) (millimeters of mercury [mmHg]): 40, 110; Systolic blood pressure (SBP) (mmHg): 90, 170; Heart rate (beats per minute): 35, 120. LLN=lower limit of normal; ULN=upper limit of normal.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 148 | 0
Participants
  DBP, TC 1, BL, <LLN, n=0, 148, 0 |  | 0 |
  DBP, TC 1, PBL, <LLN, n=0, 148, 0 |  | 2 |
  DBP, TC 1, BL, >ULN, n=0, 148, 0 |  | 0 |
  DBP, TC 1, PBL, >ULN, n=0, 148, 0 |  | 1 |
  SBP, TC 1, BL, <LLN, n=0, 148, 0 |  | 0 |
  SBP, TC 1, PBL, <LLN, n=0, 148, 0 |  | 7 |
  SBP, TC 1, BL, >ULN, n=0, 148, 0 |  | 0 |
  SBP, TC 1, PBL, >ULN, n=0, 148, 0 |  | 7 |
  HR, TC 1, BL, <LLN, n=0, 148, 0 |  | 0 |
  HR, TC 1, PBL, <LLN, n=0, 148, 0 |  | 0 |
  HR, TC 1, BL, >ULN, n=0, 148, 0 |  | 0 |
  HR, TC 1, PBL, >ULN, n=0, 148, 0 |  | 1 |
  DBP, TC 2, BL, <LLN, n=0, 93, 0 |  | 0 |
  DBP, TC 2, PBL, <LLN, n=0, 93, 0 |  | 0 |
  DBP, TC 2, BL, >ULN, n=0, 93, 0 |  | 0 |
  DBP, TC 2, PBL, >ULN, n=0, 93, 0 |  | 0 |
  SBP, TC 2, BL, <LLN, n=0, 93, 0 |  | 0 |
  SBP, TC 2, PBL, <LLN, n=0, 93, 0 |  | 3 |
  SBP, TC 2, BL, >ULN, n=0, 93, 0 |  | 0 |
  SBP, TC 2, PBL, >ULN, n=0, 93, 0 |  | 6 |
  HR, TC 2, BL, <LLN, n=0, 93, 0 |  | 0 |
  HR, TC 2, PBL, <LLN, n=0, 93, 0 |  | 0 |
  HR, TC 2, BL, >ULN, n=0, 93, 0 |  | 0 |
  HR, TC 2, PBL, >ULN, n=0, 93, 0 |  | 1 |
  DBP, TC 3, BL, <LLN, n=0, 62, 0 |  | 0 |
  DBP, TC 3, PBL, <LLN, n=0, 63, 0 |  | 0 |
  DBP, TC 3, BL, >ULN, n=0, 62, 0 |  | 0 |
  DBP, TC 3, PBL, >ULN, n=0, 63, 0 |  | 0 |
  SBP, TC 3, BL, <LLN, n=0, 62, 0 |  | 0 |
  SBP, TC 3, PBL, <LLN, n=0, 63, 0 |  | 0 |
  SBP, TC 3, BL, >ULN, n=0, 62, 0 |  | 0 |
  SBP, TC 3, PBL, >ULN, n=0, 63, 0 |  | 0 |
  HR, TC 3, BL, <LLN, n=0, 62, 0 |  | 0 |
  HR, TC 3, PBL, <LLN, n=0, 63, 0 |  | 0 |
  HR, TC 3, BL, >ULN, n=0, 62, 0 |  | 0 |
  HR, TC 3, PBL, >ULN, n=0, 63, 0 |  | 0 |
  DBP, TC 4, BL, <LLN, n=0, 29, 0 |  | 0 |
  DBP, TC 4, PBL, <LLN, n=0, 30, 0 |  | 0 |
  DBP, TC 4, BL, >ULN, n=0, 29, 0 |  | 0 |
  DBP, TC 4, PBL, >ULN, n=0, 30, 0 |  | 0 |
  SBP, TC 4, BL, <LLN, n=0, 29, 0 |  | 0 |
  SBP, TC 4, PBL, <LLN, n=0, 30, 0 |  | 2 |
  SBP, TC 4, BL, >ULN, n=0, 29, 0 |  | 0 |
  SBP, TC 4, PBL, >ULN, n=0, 30, 0 |  | 1 |
  HR, TC 4, BL, <LLN, n=0, 29, 0 |  | 0 |
  HR, TC 4, PBL, <LLN, n=0, 30, 0 |  | 0 |
  HR, TC 4, BL, >ULN, n=0, 29, 0 |  | 0 |
  HR, TC 4, PBL, >ULN, n=0, 30, 0 |  | 0 |
  DBP, TC 5, BL, <LLN, n=0, 13, 0 |  | 0 |
  DBP, TC 5, PBL, <LLN, n=0, 13, 0 |  | 0 |
  DBP, TC 5, BL, >ULN, n=0, 13, 0 |  | 0 |
  DBP, TC 5, PBL, >ULN, n=0, 13, 0 |  | 0 |
  SBP, TC 5, BL, <LLN, n=0, 13, 0 |  | 0 |
  SBP, TC 5, PBL, <LLN, n=0, 13, 0 |  | 2 |
  SBP, TC 5, BL, >ULN, n=0, 13, 0 |  | 0 |
  SBP, TC 5, PBL, >ULN, n=0, 13, 0 |  | 0 |
  HR, TC 5, BL, <LLN, n=0, 13, 0 |  | 0 |
  HR, TC 5, PBL, <LLN, n=0, 13, 0 |  | 0 |
  HR, TC 5, BL, >ULN, n=0, 13, 0 |  | 0 |
  HR, TC 5, PBL, >ULN, n=0, 13, 0 |  | 0 |
  DBP, TC 6, BL, <LLN, n=0, 6, 0 |  | 0 |
  DBP, TC 6, PBL, <LLN, n=0, 6, 0 |  | 0 |
  DBP, TC 6, BL, >ULN, n=0, 6, 0 |  | 0 |
  DBP, TC 6, PBL, >ULN, n=0, 6, 0 |  | 0 |
  SBP, TC 6, BL, <LLN, n=0, 6, 0 |  | 0 |
  SBP, TC 6, PBL, <LLN, n=0, 6, 0 |  | 1 |
  SBP, TC 6, BL, >ULN, n=0, 6, 0 |  | 0 |
  SBP, TC 6, PBL, >ULN, n=0, 6, 0 |  | 0 |
  HR, TC 6, BL, <LLN, n=0, 6, 0 |  | 0 |
  HR, TC 6, PBL, <LLN, n=0, 6, 0 |  | 0 |
  HR, TC 6, BL, >ULN, n=0, 6, 0 |  | 0 |
  HR, TC 6, PBL, >ULN, n=0, 6, 0 |  | 0 |

42. Secondary Outcome: Number of Participants With Immunoglobulin Values Outside the Reference Range at Baseline or Any Visit Post-baseline, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The baseline value for a treatment course is defined as the latest value on or before the date of infusion A of the treatment course. The post-baseline visit is defined as any visit after the date of infusion A during the specified treatment course. Reference ranges (LLN, ULN) used for immunoglobulins are: immunoglobulin A (IgA) (grams/Liter): 0.81, 4.63; immunoglobulin G (IgG) (grams/Liter): 6.94, 16.18; immunoglobulin M (IgM) (grams/Liter): 0.48, 2.71.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 141 | 0
Participants
  IgA, TC 1, BL, <LLN, n=0, 141, 0 |  | 1 |
  IgA, TC 1, PBL, <LLN, n=0, 133, 0 |  | 1 |
  IgA, TC 1, BL, >ULN, n=0, 141, 0 |  | 16 |
  IgA, TC 1, PBL, >ULN, n=0, 133, 0 |  | 14 |
  IgG, TC 1, BL, <LLN, n=0, 141, 0 |  | 0 |
  IgG, TC 1, PBL, <LLN, n=0, 133, 0 |  | 4 |
  IgG, TC 1, BL, >ULN, n=0, 141, 0 |  | 43 |
  IgG, TC 1, PBL, >ULN, n=0, 133, 0 |  | 25 |
  IgM, TC 1, BL, <LLN, n=0, 141, 0 |  | 7 |
  IgM, TC 1, PBL, <LLN, n=0, 133, 0 |  | 18 |
  IgM, TC 1, BL, >ULN, n=0, 141, 0 |  | 19 |
  IgM, TC 1, PBL, >ULN, n=0, 133, 0 |  | 12 |
  IgA, TC 2, BL, <LLN, n=0, 85, 0 |  | 0 |
  IgA, TC 2, PBL, <LLN, n=0, 93, 0 |  | 0 |
  IgA, TC 2, BL, >ULN, n=0, 85, 0 |  | 9 |
  IgA, TC 2, PBL, >ULN, n=0, 93, 0 |  | 1 |
  IgG, TC 2, BL, <LLN, n=0, 85, 0 |  | 1 |
  IgG, TC 2, PBL, <LLN, n=0, 93, 0 |  | 3 |
  IgG, TC 2, BL, >ULN, n=0, 85, 0 |  | 11 |
  IgG, TC 2, PBL, >ULN, n=0, 93, 0 |  | 12 |
  IgM, TC 2, BL, <LLN, n=0, 85, 0 |  | 10 |
  IgM, TC 2, PBL, <LLN, n=0, 93, 0 |  | 18 |
  IgM, TC 2, BL, >ULN, n=0, 85, 0 |  | 6 |
  IgM, TC 2, PBL, >ULN, n=0, 93, 0 |  | 5 |
  IgA, TC 3, BL, <LLN, n=0, 59, 0 |  | 0 |
  IgA, TC 3, PBL, <LLN, n=0, 62, 0 |  | 0 |
  IgA, TC 3, BL, >ULN, n=0, 59, 0 |  | 5 |
  IgA, TC 3, PBL, >ULN, n=0, 62, 0 |  | 5 |
  IgG, TC 3, BL, <LLN, n=0, 59, 0 |  | 0 |
  IgG, TC 3, PBL, <LLN, n=0, 62, 0 |  | 2 |
  IgG, TC 3, BL, >ULN, n=0, 59, 0 |  | 6 |
  IgG, TC 3, PBL, >ULN, n=0, 62, 0 |  | 5 |
  IgM, TC 3, BL, <LLN, n=0, 59, 0 |  | 7 |
  IgM, TC 3, PBL, <LLN, n=0, 62, 0 |  | 11 |
  IgM, TC 3, BL, >ULN, n=0, 59, 0 |  | 3 |
  IgM, TC 3, PBL, >ULN, n=0, 62, 0 |  | 2 |
  IgA, TC 4, BL, <LLN, n=0, 28, 0 |  | 0 |
  IgA, TC 4, PBL, <LLN, n=0, 29, 0 |  | 0 |
  IgA, TC 4, BL, >ULN, n=0, 28, 0 |  | 4 |
  IgA, TC 4, PBL, >ULN, n=0, 29, 0 |  | 5 |
  IgG, TC 4, BL, <LLN, n=0, 28, 0 |  | 0 |
  IgG, TC 4, PBL, <LLN, n=0, 29, 0 |  | 1 |
  IgG, TC 4, BL, >ULN, n=0, 28, 0 |  | 1 |
  IgG, TC 4, PBL, >ULN, n=0, 29, 0 |  | 1 |
  IgM, TC 4, BL, <LLN, n=0, 28, 0 |  | 1 |
  IgM, TC 4, PBL, <LLN, n=0, 29, 0 |  | 2 |
  IgM, TC 4, BL, >ULN, n=0, 28, 0 |  | 1 |
  IgM, TC 4, PBL, >ULN, n=0, 29, 0 |  | 1 |
  IgA, TC 5, BL, <LLN, n=0, 12, 0 |  | 0 |
  IgA, TC 5, PBL, <LLN, n=0, 13, 0 |  | 0 |
  IgA, TC 5, BL, >ULN, n=0, 12, 0 |  | 2 |
  IgA, TC 5, PBL, >ULN, n=0, 13, 0 |  | 2 |
  IgG, TC 5, BL, <LLN, n=0, 12, 0 |  | 1 |
  IgG, TC 5, PBL, <LLN, n=0, 13, 0 |  | 1 |
  IgG, TC 5, BL, >ULN, n=0, 12, 0 |  | 0 |
  IgG, TC 5, PBL, >ULN, n=0, 13, 0 |  | 1 |
  IgM, TC 5, BL, <LLN, n=0, 12, 0 |  | 0 |
  IgM, TC 5, PBL, <LLN, n=0, 13, 0 |  | 0 |
  IgM, TC 5, BL, >ULN, n=0, 12, 0 |  | 1 |
  IgM, TC 5, PBL, >ULN, n=0, 13, 0 |  | 1 |
  IgA, TC 6, BL, <LLN, n=0, 6, 0 |  | 0 |
  IgA, TC 6, PBL, <LLN, n=0, 6, 0 |  | 0 |
  IgA, TC 6, BL, >ULN, n=0, 6, 0 |  | 0 |
  IgA, TC 6, PBL, >ULN, n=0, 6, 0 |  | 0 |
  IgG, TC 6, BL, <LLN, n=0, 6, 0 |  | 0 |
  IgG, TC 6, PBL, <LLN, n=0, 6, 0 |  | 0 |
  IgG, TC 6, BL, >ULN, n=0, 6, 0 |  | 0 |
  IgG, TC 6, PBL, >ULN, n=0, 6, 0 |  | 0 |
  IgM, TC 6, BL, <LLN, n=0, 6, 0 |  | 0 |
  IgM, TC 6, PBL, <LLN, n=0, 6, 0 |  | 0 |
  IgM, TC 6, BL, >ULN, n=0, 6, 0 |  | 0 |
  IgM, TC 6, PBL, >ULN, n=0, 6, 0 |  | 0 |

43. Secondary Outcome: Number of Participants With Positive John Cunningham (JC) Virus Test Results at Baseline or Any Visit Post-baseline During the DB and OL Periods
Description: Blood samples were collected for analysis of plasma/white blood cell JC Virus (JCV) using the polymerase chain reaction (PCR) assay. A positive JC Virus test result indicates the presence of JC Virus.
Time Frame: From basline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 118 | 0
Participants
  TC 1, BL, n=0, 76, 0 |  | 1 |
  TC 1, PBL, n=0, 118, 0 |  | 1 |
  TC 2, BL, n=0, 45, 0 |  | 0 |
  TC 2, PBL, n=0, 81, 0 |  | 1 |
  TC 3, BL, n=0, 30, 0 |  | 1 |
  TC 3, PBL, n=0, 48, 0 |  | 0 |
  TC 4, BL, n=0, 10, 0 |  | 0 |
  TC 4, PBL, n=0, 25, 0 |  | 0 |
  TC 5, BL, n=0, 4, 0 |  | 0 |
  TC 5, PBL, n=0, 8, 0 |  | 0 |
  TC 6, BL, n=0, 3, 0 |  | 0 |
  TC 6, PBL, n=0, 6, 0 |  | 0 |

44. Secondary Outcome: Number of Participants With Any Serious Adverse Event During the Follow-up Period
Description: A serious adverse event is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; or is a congenital anomaly/birth defect. Medical or scientific judgment should have been exercised in other situations. Refer to the general SAE module for a list of SAEs.
Time Frame: From the last scheduled visit in the DB or OL Period until B-cells and circulating IgG had returned to normal or baseline levels (or maximum of 2 years from Last Subject Last Visit [LSLV])
Population: Safety Follow-up Population: all participants who withdrew from the Double-blind Period and had evidence of contact with the site after the end of the Double-blind Period and all participants who withdrew or completed the Open-label Period and had evidence of contact with the site after their end of Open-label date.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 0 | 132
Participants |  |  | 17

45. Secondary Outcome: Number of Participants With Immunoglobulin Values Outside the Reference Range During the Follow-up Period
Description: The reference ranges for immunoglobulins (LLN, ULN) are defined as: IgA (grams/Liter): 0.81, 4.63; IgG (grams/Liter): 6.94, 16.18; IgM (grams/Liter): 0.48, 2.71.
Time Frame: From the last scheduled visit in the DB or OL Period until B-cells and circulating IgG had returned to normal or baseline levels (or maximum of 2 years from LSLV)
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 0 | 123
Participants
  IgA <LLN |  |  | 0
  IgA >ULN |  |  | 15
  IgG <LLN |  |  | 7
  IgG >ULN |  |  | 18
  IgM <LLN |  |  | 23
  IgM >ULN |  |  | 4

46. Secondary Outcome: Time to First CD19+ B-cell Repopulation Relative to the First Dose and Last Dose of Ofatumumab
Description: Time to first CD19+ B-cell repopulation (return to normal or baseline level) relative to the first dose was assessed only for those participants whose B-cells repopulated after receiving ofatumumab. Time to first CD19+ B-cell repopulation relative to the last dose of ofatumumab was assessed only for those participants whose B-cells repopulated during their last ofatumumab treatment course or follow-up.
Time Frame: From the first dose of ofatumumab until the last Follow-up Period visit (up to Week 248)
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Median (Full Range); unit: Months
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 0 | 63
Months
  Relative to first dose, n=0, 0, 63 |  |  | 22.013 [0.46 to 49.25]
  Relative to last dose, n=0, 0, 60 |  |  | 12.567 [0.03 to 29.47]

47. Secondary Outcome: Number of Participants With a Positive JC Virus Test Result During the Follow-up Period
Description: Blood samples were collected for analysis of plasma/white blood cell JC Virus (JCV) using the polymerase chain reaction (PCR) assay. Positive JC Virus test result indicated presence of JC Virus.
Time Frame: as for outcome 45
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 0 | 132
Participants |  |  | 7

48. Secondary Outcome: Number of Participants With the Indicated Clinical Chemistry Values of Potential Clinical Concern During the Follow-up Period
Description: Only those parameters for which at least one value of clinical concern (CC) was reported are summarized. Pre-defined limits of potential clinical concern (CC Low [relative to the lower limit of normal], CC High [relative to the upper limit of normal]) are: ALT: NA, 2; ALP: NA, 1.5; TBIL: NA, 1.5; CO2/BCO: 0.85, 1.2; CK: NA, 2; GGT: NA, 2; Urea/BUN: NA, 1.5.
Time Frame: From the last scheduled visit in the DB or OL Period until B-cells and circulating IgG had returned to normal or baseline levels (maximum of 2 years)
Population: AT Population. Only participants who withdrew from the DB Period and had evidence of contact with the site after the end of the DB Period and all participants who withdrew or completed the OL Period and had evidence of contact with the site after their end of OL date were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 0 | 132
Participants
  ALT |  |  | 1
  ALP |  |  | 1
  CK |  |  | 2
  CO2/BCO |  |  | 2
  GGT |  |  | 1
  TBIL |  |  | 1
  Urea/BUN |  |  | 1

49. Secondary Outcome: Number of Participants With the Indicated Hematology Values of Potential Clinical Concern During the Follow-up Period
Description: Only those parameters for which at least one value of clinical concern (CC) was reported are summarized. Pre-defined limits of potential clinical concern (CC Low [relative to lower limit of normal], CC High [relative to upper limit of normal]) are: Eosinophils: NA, 2; Total neutrophils: 0.8, 1.6; Platelet count: 0.65, 1.5.
Time Frame: as for outcome 48
Population: as for outcome 48
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 0 | 132
Participants
  Eosinophils |  |  | 1
  Total neutrophils |  |  | 2
  Platelet count |  |  | 1

ADVERSE EVENTS:
Time Frame: Because no investigational product was administered during the Follow-up Period, per protocol, only serious adverse events (SAEs) were collected and reported for this period.
Description: SAEs/AEs were collected in members of the Safety Population (SP), which is identical to the ITT Population, except that participants were analyzed according to the actual treatment received rather than to the treatment randomized to (one participant was randomized to placebo but received study drug).
Groups:
- Placebo: DB Period: Serious adverse events (SAEs) and non-serious AEs are reported for participants receiving placebo in the DB Period. Placebo was administered as two 1000 milliliter (ml) intravenous (IV) infusions, one at Day 0 and the other at Day 14, in addition to background methotrexate (MTX) treatment (7.5 to 25 milligrams [mg]/week [oral, intramuscular, or subcutaneous] for 24 weeks) in the DB Period.
- Ofatumumab 700 mg: DB and OL Periods: SAEs and non-serious AEs are reported for participants receiving ofatumumab 700 mg in either the DB or OL Period. Ofatumumab 700 mg (35 ml) was administered as two 1000 ml IV infusions, one at Day 0 and the other at Day 14, in addition to background MTX treatment (7.5 to 25 mg/week [oral, intramuscular, or subcutaneous] for 24 weeks) in the DB Period. Participants completing the 24-week DB Period without receiving rescue disease-modifying anti-rheumatic drug treatment were eligible to proceed into the 120-week OL Period to receive repeat ofatumumab treatment courses (at individualized time intervals if a clinical response had been achieved after the previous treatment course).
- Placebo or Ofatumumab 700 mg: Follow-up Period: SAEs and non-serious AEs are reported for participants receiving either placebo or ofatumumab 700 mg in the Follow-up Period. Participants randomized to DB treatment who completed the OL Period, who did not enter the OL Period, who did not qualify for retreatment, or who were withdrawn were to be followed until the number of B-cells and circulating IgG had returned to normal (according to the central laboratory) or Baseline levels or for a maximum of 2 years from the last scheduled visit in the DB or OL Periods, whichever occurred earlier. No investigational product was administered in the Follow-up Period.
Arm/Group | Placebo: DB Period | Ofatumumab 700 mg: DB and OL Periods | Placebo or Ofatumumab 700 mg: Follow-up Period
Serious Adverse Events (participants affected / at risk) | 6/83 | 30/148 | 17/132
Other Adverse Events (participants affected / at risk) | 36/83 | 133/148 | 0/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: DB Period (N=83) | Ofatumumab 700 mg: DB and OL Periods (N=148) | Placebo or Ofatumumab 700 mg: Follow-up Period (N=132)
Anaphylactic reaction (Immune system disorders) | 0 | 4 | 0
Hypersensitivity (Immune system disorders) | 0 | 2 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0
John Cunningham (JC) virus test positive (Investigations) | 1 | 0 | 2
Cervical myelopathy (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Herpes oesophagitis (Infections and infestations) | 0 | 1 | 0
Implant site reaction (General disorders) | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Haemophilus infection (Infections and infestations) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intervertebral disc protrusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: DB Period (N=83) | Ofatumumab 700 mg: DB and OL Periods (N=148) | Placebo or Ofatumumab 700 mg: Follow-up Period (N=132)
Rash (Skin and subcutaneous tissue disorders) | 2 | 53 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 16 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 19 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 24 | 0
Gastroenteritis (Infections and infestations) | 4 | 9 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 20 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 9 | 0
Nasopharyngitis (Infections and infestations) | 5 | 7 | 0
Urinary tract infection (Infections and infestations) | 4 | 9 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 7 | 0
Dizziness (Nervous system disorders) | 0 | 8 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 13 | 0
Headache (Nervous system disorders) | 3 | 4 | 0
Nausea (Gastrointestinal disorders) | 2 | 5 | 0
Rhinitis (Infections and infestations) | 2 | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 4 | 0
Blood pressure increased (Investigations) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Pyrexia (General disorders) | 2 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 6 | 0
Alanine aminotransferase increased (Investigations) | 0 | 5 | 0
Cervicitis (Infections and infestations) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 6 | 0
Dry eye (Eye disorders) | 2 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Flushing (Vascular disorders) | 0 | 6 | 0
Herpes zoster (Infections and infestations) | 2 | 5 | 0
Hypertension (Vascular disorders) | 0 | 8 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 3 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Pharyngitis (Infections and infestations) | 2 | 3 | 0
Sensation of foreign body (Gastrointestinal disorders) | 0 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 10 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 8 | 0
Depression (Psychiatric disorders) | 0 | 6 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0
Anxiety (Psychiatric disorders) | 0 | 5 | 0
Cataract (Eye disorders) | 0 | 5 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Chest discomfort (General disorders) | 0 | 4 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Chest pain (General disorders) | 0 | 3 | 0
Erysipelas (Infections and infestations) | 0 | 3 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 3 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Sciatica (Nervous system disorders) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.